# **Statistical Analysis Plan for:**

Study IMM-101-008 NCT01559818

A Long Term Follow up Study for Patients Who Previously Took Part in the Phase I Study IMM-101-001

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

**Customer:** Immodulon Therapeutics Limited **Information Type:** Statistical Analysis Plan

| Title: | Statistical Analysis Plan for IMM-101-008 (long-term follow-up [LTF] study) |
|---|---|
| Version | Amendment 1 |
| Effective Date: | 10 April 2019 |

**Description:** An open label long-term follow-up study of patients with melanoma who were previously enrolled in the Phase I study IMM-101-001 (first-in-human [FIH] study).

Author's Name, Title and Functional Area: Sarah Taggart, Statistician, Exploristics Ltd

Helen Amine-Eddine, Consultant Statistician, KataCliniKa Ltd

Moira Murphy, Statistician, Exploristics Ltd

Approved by:

Helen Amine-Eddine

Consultant Statistician, KataCliniKa Ltd on behalf of Immodulon Therapeutics Ltd

Helen Amine-Eddine

Ma- Ma. A

Moira Murphy

Statistician Exploristics Ltd 10 April 2019

\_\_\_\_

10 Apr2019

Date

Copyright 2019 Exploristics Limited. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

| Audit Trail For This Document | | | |
|---|---|---|---|
| Compiled by/Affiliation | Type of Change | Date | Version |
| Sarah Taggart | Creation | 06 January 2015 | 0.1 |
| Anne-Marie Duggan | Internal review | 18 February 2015 | 1.0 |
| Immodulon | Review | 28 April 2015 | 1.1 |
| Sarah Taggart | Updates based on clients' comments | 08 May 2015 | 2.0 |
| Sarah Taggart | Updates based on client TC (18 MAY 2015) | 28 May 2015 | 3.0 |
| Immodulon | Review | 12 June 2015 | 3.1 |
| Sarah Taggart | Updates based on client review and correspondence | 26 June 2015 | 3.2 |
| Anne-Marie Duggan | Internal review | 01 July 2015 | 3.3 |
| Sarah Taggart | Pre-Final Draft | 09 July 2015 | Pre-Final Draft |
| Immodulon | Review | 16 September<br>2015 | Final Draft 1 |
| Sarah Taggart | Updates following client review | 30 September<br>2015 | Final Draft 2 |
| Anne-Marie | Final internal review | 06 October 2015 | Final Review |
| Sarah Taggart | Updates following final review | 07 October 2015 | Final |
| Effective Date | | 08 October 2015 | Final |
| Immodulon | Updates following review of SAP prior to final database lock and including relevant tables including IMM-101-001 and IMM-101-008 data for the Safety population of IMM-101-008 study, from the retired SAP Addendum. | 28 January 2019 | Amendment 1,<br>Draft 1 |
| Exploristics Ltd | Review | 11 February 2019 | Amendment 1,<br>Draft 1 |
| Immodulon | Incorporation of clarifications received following Exploristics review and Immodulon review comments | 11 February 2019 | Amendment 1,<br>Draft 2 |
| Exploristics Ltd | Final internal review | 14 March 2019 | Amendment 1,<br>Draft 3 |
| Clare Gleeson | Review (incorporating review by Exploristics Ltd) | 14 March 2019 | Final Draft |
| Effective Date | Incorporation of review comments and approval | 10 April 2019 | Final Amendment 1 |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

# **Table of Contents**

| ABBREVIATIONS | 4 |
|--------------------------------------------------------------|----|
| 1. INTRODUCTION | 5 |
| 2. STUDY OBJECTIVE(S) AND ENDPOINT(S) | 6 |
| 2.1 Study Objective(s) | 6 |
| 2.2 Study Endpoint(s) | 6 |
| 3. STUDY DESIGN | 7 |
| 4. PLANNED ANALYSES | 7 |
| 5. SAMPLE SIZE CONSIDERATIONS | 8 |
| 6. ANALYSIS POPULATIONS | 8 |
| 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES | 8 |
| 8. DATA HANDLING CONVENTIONS | 9 |
| 8.1 Premature Withdrawal and Missing Data | 9 |
| 8.3 Derived and Transformed Data | 10 |
| 9. DESCRIPTIVE STATISTICS | 13 |
| 9.1 Disposition of Patients | 13 |
| 9.2 Demographic and Baseline Characteristics | 13 |
| 9.3 Study Treatment, Exposure and Safety Outputs | 13 |
| 10. ANALYSIS CORRESPONDING TO THE STUDY OBJECTIVES | 15 |
| 11. PROTOCOL DEVIATIONS AND DEVIATIONS FROM PLANNED ANALYSIS | 16 |
| 12. REFERENCES | 16 |
| 13. ATTACHMENTS | 17 |
| 13.1 Table of Contents for Data Display Specifications | 17 |
| 13.2 Data Display Specification | 19 |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

# **ABBREVIATIONS**

| ADaM | Analysis Data Model |
|---------|------------------------------------------------------------|
| | Analysis Data Model |
| AE | Adverse Event |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| FIH | First-in-human |
| LTF | Long-term follow-up |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| NCI | National Cancer Institute |
| NPP | Named Patient Programme |
| OS | Overall Survival |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TFL | Tables, Figures and Listings |
| Yrs | Years |

Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

#### 1. INTRODUCTION

The study explores the long-term safety and tolerability of continued administration of IMM-101 in patients who were previously enrolled in the Phase I safety and tolerability study, IMM-101-001. IMM-101-001 was a first-in-human (FIH), open-label, dose-escalation, intra-patient, placebo-controlled study, in adult patients with confirmed diagnosis of stage III or IV melanoma to evaluate the safety and tolerability of three doses of IMM-101 (further details are available in the FIH study clinical study report [CSR]).

In this long-term follow-up (LTF) study, IMM-101-008, IMM-101 (10 mg/mL) is administered as a single 0.1 mL intradermal injection every 4 weeks or as close to this interval as permitted due to practical or logistical considerations until death or withdrawal, unless such therapy is contraindicated, the patient does not wish to continue, or the study is terminated by the Sponsor.

The duration of this study is determined by the time to death or withdrawal of the last patient remaining in this study, hence the total duration of the study is not pre-determined.

This Statistical Analysis Plan (SAP) describes the intended statistical evaluation of the study data at the time of final study reporting based on the final study database.

This SAP is based on the study protocol (version 9.0, dated 18 October 2017, incorporating amendment numbers 1.0 to 8.0) and the final study case report form (CRF), version 4, dated 02 December 2012, the amended adverse event (AE) CRF version 3, dated 15 October 2013, and Post-Study Long Term Survival Status CRF version 1.0, dated 28 September 2015.

This SAP incorporates the original objectives outlined in the study protocol, the approved SAP dated 08 October 2015 and further amendments combining relevant data from the FIH study IMM-101-001 with the final study data for the LTF study IMM-101-008, in IMM-101-008-enrolled patients, thus providing an evaluation of the long-term safety profile of IMM-101 from first dosing in the FIH study through to last dosing in the LTF study, including the period between studies when patients were treated with IMM-101 under the Immodulon Named Patient Programme (NPP), when relevant data has been recorded in the LTF study CRF.

The FIH study results are reported in the CSR (date 01 March 2011), based on the final FIH study CRF version date 25 January 2010 and the final study database.

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

# 2. STUDY OBJECTIVE(S) AND ENDPOINT(S)

### 2.1 Study Objective(s)

The study objectives are,

- To determine the long-term safety profile of IMM-101 administered intradermally for extended use.
- To document the long-term clinical course of the patients previously enrolled in Study IMM-101-001.
- To monitor selected markers of tumour burden and immunological status.

The objective of this Statistical Analysis Plan (SAP) is to summarise the following outputs:

- Patient disposition
- Demographic characteristics
- Medical history
- Previous medications
- IMM-101 dose administration, time on study and exposure
- Injection site reactions
- Adverse events
- Overall Survival (OS)

The FIH and LTF combined data presentation objectives are to summarise the following outputs:

- Relevant medical events during the NPP (i.e. prior to entry to IMM-101-008)
- Anti-melanoma Cancer Therapies other than IMM-101 whilst on IMM-101 treatment
- IMM-101 administrations (from first dose of IMM-101 in the FIH study and including administrations during the LTF study)
- IMM-101 exposure
- Incidence and frequency of IMM-101-related treatment emergent AEs occurring following first dose
  of IMM-101 in the FIH study

# 2.2 Study Endpoint(s)

The Safety and Tolerability endpoints are:

- Local injection site tolerability
- Adverse Events with documentation of number, type and degree of toxicities as measured by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) v4.0 [1] where appropriate.

The Efficacy endpoints are:

- Overall survival
- Reduction in metastatic disease.

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Exploratory endpoints of change in markers of immune status are to be reported separately from the main endpoints of the study, and the analyses are not therefore described in this SAP.

### 3. STUDY DESIGN

The LTF study is an open label long-term follow-up study of patients with melanoma who were previously enrolled in the Phase I FIH study IMM-101-001. The study consists of two phases; screening and enrolment, then treatment.

The screening period lasted up to 28 days to establish eligibility. Once confirmed as eligible, patients receive treatment every 4 weeks or as close to this interval as is permitted due to practical or logistical considerations until death or withdrawal, unless such therapy is contraindicated, the patient does not wish to continue or the study is terminated by the Sponsor. The dose interval can be modified at the discretion of the Investigator provided the minimum period between doses is no less than 14 days.

IMM-101 can be stopped if deemed necessary by the Investigator and/or patient, for example, due to intolerable injection site reactions. In the event of an injection site reaction of Grade 3 and above, at the discretion of the Investigator, patients may be administered a half dose of the study drug (i.e., a single 0.05 mL intradermal injection of IMM-101) or the time interval between doses may be increased. Patients can choose to withdraw from the study at any time and for any reason.

Protocol amendment 6.0 (dated 07 November 2014) allowed for a clinic telephone call to the patient to enquire about injection site reactions, adverse events, concomitant medications and any other concerns, if the patient does not attend for a study visit within a calendar month. Appropriate information is recorded in the CRF.

#### 4. PLANNED ANALYSES

At the time of final analysis for the study, descriptive summaries of the results of the study will be provided along with data listings of the final study database. Summary statistics or frequency tables will be provided, where appropriate.

Section 9 provides details of the descriptive statistics and TFL shells are included in Section 13.

No formal statistical analyses of the results are anticipated and hence no statistical inferences will be made.

Planned analyses as detailed in the protocol are as follows:

The evaluation of safety and tolerability will be summarised using the Safety population and will be based on local and systemic toxicities (including injection site tolerability) which will be presented over the treatment period in standard frequency tables, overall and by number, degree and type. Adverse Events will

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

be presented descriptively to include related adverse events, serious adverse events (SAEs), and adverse events leading to withdrawal or death. The frequency and severity of injection site reactions, and all other safety parameters will be summarised.

All patients will have received IMM-101 in the context of both the Phase 1 study and, for the majority, on a Named Patient basis; therefore all AEs in this long term follow up study will be regarded as treatment emergent.

Efficacy will be presented using the Safety population and will be assessed through documenting the long-term clinical course of the patients previously enrolled in Study IMM-101-001 in terms of OS. Reduction in metastatic disease will be listed only.

Variables for the exploratory endpoints will be analysed and reported separately to the main efficacy and safety endpoints of the study.

The protocol specified that OS will be presented from enrolment into this study, in addition to time from initial diagnosis and enrolment into study IMM-101-001. Time zero for the OS analysis in this study (IMM-101-008) will be based on the date of Day 0 in this study and analysis of OS taking into account time from initial diagnosis and first dosing day in Study IMM-101-001 will not be included in this SAP as not all patients completing the FIH study entered the LTF study.

In addition to the above planned presentations, non-serious adverse events in LTF study patients will be tabulated and treatment-related treatment emergent AEs will also be presented combining data in these patients, from both the FIH and LTF studies.

### 5. SAMPLE SIZE CONSIDERATIONS

Surviving patients from Study IMM-101-001 (EudraCT number: 2009-012447-42) who were continuing to receive IMM-101 on a Named Patient Programme (NPP) basis were invited to enrol into study IMM-101-008.

#### 6. ANALYSIS POPULATIONS

The Safety Population will comprise all patients who receive at least one dose of the study drug in the LTF study. All members of the Safety Population had previously been enrolled into the FIH study. Analysis of safety and tolerability endpoints and efficacy endpoints will be summarised on the Safety Population.

#### 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES

In general, continuous data will be summarised using mean, standard deviation, minimum, median and maximum. The minimum and maximum will be recorded to the same number of significant figures as the

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

original data, whilst mean and median will be presented to 1 significant figure more than the original data, and standard deviation 2 significant figures more than the original data.

In summaries of categorical data, frequency counts and percentages will be used. Generally, percent will be displayed to one decimal place.

The time to event variable OS will be analysed using standard Kaplan-Meier techniques. The Kaplan Meier curve will be plotted and median (50%), 25% and 75% survival estimates reported with the corresponding 95% confidence intervals (CIs).

All analyses will be performed using SAS v 9.4 (or higher).

All tables, figures and listings (TFLs) will include titles, headers or footnotes which identify:-

- The analysis set on which the presentation is based.
- A description or title for the presentation (where combined data is presented from the FIH study and the LTF study, this will be indicated).
- The date and time the output was produced.
- A reference to the name and location of the file used to produce the output and the source of the data used (which may be a SAS dataset or another TFL).
- Reference to the analysis stage of the study data e.g. Final Analysis.

Listings which present data using repeating rows for a patient and/or visit will be presented in chronological date order (where applicable) with the repeating header information presented on the first new record for each repeating combination only, to facilitate readability.

All assessment data will be reported with the visit at which it was recorded, whether or not the visit falls inside the relevant window or not.

Tables and figures will be coded from Analysis Data Model (ADaM) format datasets. Listings will be coded from Study Data Tabulation Model (SDTM) datasets.

#### 8. DATA HANDLING CONVENTIONS

### 8.1 Premature Withdrawal and Missing Data

Patients who withdraw early will be included in the analysis of safety and efficacy. Missing, unused and spurious data will be treated as such. No imputation methods will be applied, except for concomitant medication stop date as follows:

If the stop date for a medication is partially missing, it will be assumed to be a concomitant medication if, based on the partial information available, concomitant is not ruled out. Hence the date will be imputed to the end of the month/year, i.e. if day is unknown it will be set to the last day of the specified month, if day S:\Services\Immodulon\IMM-101-008\SMF\SAP\IMM-101-008\_SAPvFinal 1.1


**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

and month are unknown it will be imputed as 31<sup>st</sup> December. This imputation will be also used in the determination of whether the previous medication was stopped within 14 days prior to Day 0.

Date imputations will not be shown in data listings however, the flag based on imputed dates will be shown in the listings. Date imputations will be incorporated into tabulations of previous/concomitant medications.

## 8.2 Prior and Concomitant Therapy and Medical History Melanoma Therapies Coding

Each concomitant therapy recorded during the FIH and LTF studies will be categorised according to antimelanoma cancer therapy type as follows:

Chemotherapy

Cancer surgery (note: melanoma cancer surgeries only are included in this category)

Radiotherapy

Immunotherapy (other than IMM-101)

Radiofrequency ablation

Immunotherapy IMM-101.

Other categories may be considered, if relevant and mutually exclusive to the above.

A look-up table will be created containing the relevant verbatim term, dataset location and therapy code. Exploristics will supply dataset(s) in Excel format where verbatim terms for therapies contained in the previous and concomitant medications, and medical history datasets are listed, for allocation to one of the anti-melanoma cancer therapies codes by Immodulon. These will be medically reviewed by Immodulon and approved prior to issue of final TFLs. Listings will include the assigned categories, where allocated.

All concomitant therapy groupings with the exception of immunotherapy IMM-101 will be included in the tabulation of anti-cancer (melanoma-related) therapies. Therapies included will be all therapies given after first dose of IMM-101 in the FIH study, including co-medication during NPP treatment (recorded as medical history since leaving the FIH study) and during the LTF study.

### 8.3 Derived and Transformed Data

As age was not collected it will be derived using the patient's date of birth and date of consent. The derivation will be

Age (years) = integer part of ((patient informed consent date - date of birth + 1)/365.25).

Note that the full date of birth will be used in the calculation, but only year of birth will be listed. Patient initials will not be listed.

# **Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Time since initial diagnosis of current presentation, time since excision of primary lesion, time since excision of sentinel node and time since regional lymph node resection will be derived in years as follows;

Time since initial diagnosis of current presentation (years) = (Day 0 - date of initial diagnosis of current presentation + 1)/ 365.25

Time since excision of primary lesion (years) = (Day 0 - date of excision of primary lesion + 1)/365.25.

Time since excision of sentinel node (years) = (Day 0 - date of excision of sentinel node + 1)/365.25 and missing if not excised.

Time since regional lymph node resection (years) = (Day 0 - date of regional lymph node resection + 1)/365.25 and missing if not resected.

The relevant time variable above will be reported to 1 decimal place, but calculated using all accuracy available in the data. If any dates are partial, i.e. day number missing, the time variable will be calculated using month and year only and if day and month missing, the time variable will be calculated using year only as follows:

- If only month and year are present (MMYYYY): Time since Event = (Day 0 Event date +1) / 365.25;
- If only year is present (YYYY): Time since Event = (Day 0 Event date) +1 / 365.25.

The total number of pre-study doses of IMM-101 received (since the completion of study IMM-101-001) will be calculated for each patient.

Exposure during the IMM-101-008 study will be summarised by time on study in years and overall exposure in months, which will be derived using:

**Time on study (years)** = (date of study completion (i.e. death on study)/date of withdrawal) - Day 0 + 1/365.25.

Overall study drug exposure (months) = (date of last dose - date of first dose in study IMM-101-008 + 1)/30.4375.

Overall exposure of IMM-101 (FIH and LTF study combined) will be derived using: (date of last dose in study IMM-101-008 – date of first dose in study IMM-101-001 + 1)/30.4375.

On-study dosing will be summarised using the total number of doses on study:

**Total no. doses on study** = (Total number of IMM-101 doses whilst on the LTF study by totalling the doses (full or part doses counted as 1 dose) recorded in the CRF.

Time elapsed since previous dose (for on-study administration of IMM-101) will be derived using;

S:\Services\Immodulon\IMM-101-008\SMF\SAP\IMM-101-008 SAPvFinal 1.1


**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

**Time elapsed since previous dose (days)** = (date of current dose - date of previous dose + 1).

A **dose change flag** (Dose changed from previous dose, I = increased, D = decreased) will be used to record any escalation or reduction in dose received between consecutive visits. If the dose has remained consistent compared to previous dose, this flag will remain unoccupied.

Time to event analysis will be performed on OS which will be calculated in years, from Day 0 in study IMM-101-008 using;

Overall Survival (years) = (date of death - Day 0 + 1)/365.25OR (censored date - Day 0 + 1)/365.25

See Section 10 for additional information.

Adverse events and medical history will be coded using MedDRA v 18.0 (or higher). MedDRA will be used to create System Organ Class (SOC) and Preferred Term (PT) variables.

A flag (Stopped >14 days prior) will be created for previous medications which were taken and stopped before 14 days prior to the end of screening procedures (i.e. Day 0) based on the medication end date and date of Day 0.

Previous and concomitant medications and significant medical history since completing the FIH study will undergo coding for anti-melanoma cancer treatments, see Section 8.2.

Note: Derived variables recorded in the unit of months or years will be reported to 1 decimal place, derived variables recorded in the unit of days will be reported to whole numbers only. Age will be reported to whole years only.

Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

#### 9. DESCRIPTIVE STATISTICS

### 9.1 Disposition of Patients

The number and percentage of patients meeting all inclusion criteria, completing (i.e. dying) and withdrawing will be summarised (Table 1), along with reasons for death and withdrawal from study.

### 9.2 Demographic and Baseline Characteristics

Patient demographics will be presented in Table 2.

Specific melanoma medical history is summarised in Table 3a which includes a summary of any lesions present during the screening period, by location. The number and percentage of patients with significant medical history (non-melanoma specific) since completion of study IMM-101-001 categorised by SOC and PT using MedDRA v 18.0 (or higher) will be presented in Table 3b.

Data summaries of pre-study administration by IMM-101 dose received since completing study IMM-101-001 can be found in Table 4. Pre-existing injection site reactions, and any history of severe local reactions following previous administration(s) of IMM-101 will be summarised as a frequency table (Table 5).

Previous medications are prescription/non-prescription drugs, vitamins, drugs of abuse and dietary supplements taken and stopped within 14 days prior to Day 0. Any previous medications stopped before 14 days prior to Day 0 will be identified with a flag in the listings. Any medications, including vitamins, and dietary supplements ongoing or started on/after Day 0 and surgical procedures are defined as Concomitant Therapies.

The incidence of patients receiving at least one anti-melanoma cancer therapy other than IMM-101 and ongoing or started on or after the first dose of IMM-101 in the FIH study will be summarised for the FIH and LTF studies combined. Overall incidence will be summarised as well as by therapy type and therapy verbatim term (i.e. description of treatment given). IMM-101 treatments and non-melanoma cancer therapies will not be included in the tabulation (Table 6). Concomitant treatments received during the FIH study were recorded in the FIH study CRF. Treatments for relevant medical history including relevant radiotherapy, cancer surgery, chemotherapy and immunotherapy received following completion of the FIH study and prior to entry to the LTF study and any medications taken within 14 days prior to the LTF study screening visit as well as concomitant treatments received after entry to the LTF study are recorded in the LTF study CRF.

#### 9.3 Study Treatment, Exposure and Safety Outputs

An on-study administration table (Table 7) will show the number and percentage of patients who receive study drug and whether full dose or reduced dose was administered, summarised by visit. In these

# Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

presentations, the denominator for the calculation of percentages at each visit will be based on the number of patients available at each visit who provide a response.

A line graph for each patient will be plotted to visually display any variation in doses of IMM-101 (in mg) by time, during the LTF study. This will be presented in the form of a panel plot (Figure 1a) on standard axes for each patient. Each dose will be marked by an 'X' on the plot. In addition, a panel plot (Figure 1b) will be presented including all IMM-101 doses received from the first dose in the FIH study, to the last dose in the LTF study, inclusive including those taken whilst the patient was being treated in the NPP, in a similar manner.

Exposure, to include the time on LTF study in years, overall LTF study drug exposure (months) and total no. doses on study, will be summarised in Table 9a.

Overall exposure to IMM-101 from first dose in the FIH study to last dose in the LTF study inclusive will be summarised in Table 9b.

Summaries of adverse events will include the number of adverse events and the proportion of patients experiencing at least one adverse event. If an individual patient has more than one AE at a given level of classification the patient will be counted only once at the given level of classification but each event will be counted within the number of events associated with that level of classification.

All patients will have received IMM-101 in the context of both the Phase 1 study IMM-101-001, and, for the majority, during the NPP; therefore all AEs in this long-term follow-up study will be regarded as treatment-emergent.

Table 10a includes the incidence and frequency of all TEAEs, treatment emergent treatment-related AEs, treatment emergent SAEs, Serious treatment-related TEAEs, TEAEs resulting in withdrawal or death and AEs of NCI CTCAE Grade ≥ 3.

Frequency summaries of treatment emergent adverse events by SOC and PT using MedDRA v 18.0 (or higher) will be included overall (Table 10b) and repeated to capture:-

- Treatment emergent adverse events of NCI Grade ≥3 (Table 10c)
- Treatment emergent, IMM-101-related, adverse events: AEs that are definitely, probably or possibly related to study drug or with an unknown relationship (Table 10d)
- Treatment emergent, SAEs (Table 10e)
- Treatment emergent adverse events leading to withdrawal or death (Table 10f).
- Treatment emergent non-serious adverse events (Table 10g).

Additionally, long term safety will be evaluated by combining treatment related adverse event experience in the FIH study through to the end of the LTF study by summarising treatment emergent treatment-related adverse events (IMM-101-001 and IMM-101-008 Combined) (Table 10h).

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Where it is not applicable to grade an AE using NCI CTCAE grade, it will be excluded from the summary of NCI Grade 3 and above AEs. Any AEs with missing grades, however, will be included, based on a worst-case approach.

On-study injection site reactions are summarised over the treatment period by visit in Table 11.

Urine Pregnancy Test Results and blood samples for immunological markers will be listed but not summarised.

All safety data will be listed.

Any comments recorded as free text in the CRF will be listed.

#### 10. ANALYSIS CORRESPONDING TO THE STUDY OBJECTIVES

Overall Survival (OS) is defined as the time from a patient's date of Day 0 until date of death. Patients still alive will be censored at withdrawal from the study or at last known date alive if later (where patients have consented to follow-up for overall survival outcome, after they have withdrawn from the study). If consent has been provided by the patient, the patient's final outcome will be included if death and if alive, the patient will have censored outcome at the date last known to be alive.

Post-study survival status after withdrawal from the study, for any withdrawn patients, will be recorded on a separate Post-study Long Term Survival Status CRF, and these data will be included in the analysis and data listings, as described above.

The patient's death is recorded as the date of study completion on CRF page 18 and if after withdrawal from the study, the date of death recorded on the Post-study CRF.

A patient without a death date will be censored in the analysis at the last date known to be alive providing their consent was obtained. Patients withdrawing from the study without consent for further follow up will be censored for survival at the date of their withdrawal from the study (recorded on CRF page 18).

Overall Survival will be summarised by Kaplan-Meier curves. Median, 25% and 75% survival estimates as well as associated 95% CIs will be reported in Table 8 and Figure 2.

SAS procedure output for the OS analysis will be included as an appendix to the CSR.

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

The changes in metastatic disease compared with previous assessment (as measured via CT or MRI scan) recorded at the discretion of the investigator, will be presented over the treatment period in data listings only (Listing 11).

### 11. PROTOCOL DEVIATIONS AND DEVIATIONS FROM PLANNED ANALYSIS

Protocol deviations will be reported separately, based on the study protocol deviations log maintained by Immodulon, and included in the CSR directly.

Any substantive deviations from the planned data presentations and analysis described in this SAP will be documented along with reason for change, in the CSR.

Overall survival will be calculated from the date of Day 0, not enrolment into the study, as the enrolment period may be up to 28 days long.

#### 12. REFERENCES

[1] Cancer Therapy Evaluation Program, Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0, DCTD, NHI, DHHS, 28 May 2009.

Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

# 13. ATTACHMENTS

# 13.1 Table of Contents for Data Display Specifications

| Tables | |
|---|---|
| 1 | Summary of Patient Disposition |
| 2 | Demographics |
| 3a | Melanoma Specific Medical History |
| 3b | Significant Medical History since Completion of Study IMM-101-001 |
| 4 | Pre-study IMM-101 Administration Since Completion of Study IMM-101-001 |
| 5 | Pre-Existing Injection Site Reaction(s) |
| 6 | Summary of Anti-melanoma Cancer Therapies other than IMM-101 Whilst on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined) |
| 7 | On-Study IMM-101 Administration |
| 8 | Overall Survival |
| 9a | Exposure |
| 9b | Time on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined) |
| <b>10</b> a | Summary of Treatment Emergent Adverse Events |
| 10b | Treatment Emergent Adverse Events |
| <b>10</b> c | Treatment Emergent Adverse Events with NCI CTCAE Grade ≥ 3 |
| <b>10</b> d | Treatment Emergent Adverse Events Related to IMM-101 |
| <b>10</b> e | Treatment Emergent Serious Adverse Events |
| 10f | Treatment Emergent Adverse Events Leading to Withdrawal or Death |
| 10g | Treatment emergent Non-serious Adverse Events |
| 10h | Treatment-related Treatment Emergent Adverse Events (IMM-101-001 and IMM-101-008 Combined) |
| 11 | On-Study Injection Site Reaction(s) |

| | • | | | |
|---|-----|-----|---|----|
| | | • | n | gs |
| L | .13 | SLI | | 23 |

| 1 | Patient Disposition |
|------|-----------------------------------------------------------------------|
| 2 | Demographics |
| 3a | Inclusion/Exclusion Questions |
| 3b | Inclusion/Exclusion Criteria |
| 3c | Inclusion/Exclusion Criteria Confirmation |
| 4ai | Melanoma Specific Medical History |
| 4aii | Melanoma Specific Medical History Continued |
| 4b | Significant Medical History since Completion of Study IMM-101-001 |
| 5 | Pre-Existing Injection Site Reaction(s) Assessed at Screening |
| 6 | Screening Urine Pregnancy Test Results |
| 7 | Disease and Treatment History at Screening |
| 8a | Previous Medications |
| 8b | Concomitant Therapies |
| 9 | Previous IMM-101 Administration Since Completion of Study IMM-101-001 |
| 10 | On-Study IMM-101 Administration |
| 11 | On-Study Disease Assessment |

**Exploristics Limited** 

2

#### Clinical Study Identifier: IMM-101-008 **Adverse Events** 12 On-Study Injection Site Reaction(s) 13 Concomitant Medication and Adverse Event Checks 14 Study Visits and Visit Checklists 15 Blood Sample for Immunological Markers 16 Post-Study Long Term Survival Status **17** Additional Comments Recorded 18 **Figures** Panel Plot of On-Study IMM-101 Doses by Patient **1**a All IMM-101 Dosing Administrations (IMM-101-001 and IMM-101-008 Combined) 1b

Kaplan Meier Curve of Overall Survival

Identifier: EXP12002

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

(응)

N = xx

## 13.2 Data Display Specification

Final Analysis

Protocol: IMM-101-008

Analysis Population: All patients

Page x of y

# Table 1 Summary of Patient Disposition

| | 1/1 — XX | ( 0 ) |
|---|---|---|
| Number of patients who entered the study | XX | |
| Number of patients in the safety population | XX | (xx.x) |
| Number of patients who met all Inclusion/Exclusion criteria | XX | (xx.x) |
| Number of patients who died on study | XX | (xx.x) |
| Reason for death | | |
| Adverse event/unacceptable toxicity | XX | (xx.x) |
| Other: Death due to disease progression | XX | (xx.x) |
| Number of patients who withdrew from the study | XX | (xx.x) |
| Reason for Withdrawal | | |
| Adverse event/unacceptable toxicity | XX | (xx.x) |
| Patient request/withdrawal of consent | XX | (xx.x) |
| Investigator decision | XX | (xx.x) |
| Did not meet inclusion/exclusion criteria | XX | (xx.x) |
| Pregnancy | XX | (xx.x) |
| Non-compliant | XX | (xx.x) |
| Other | XX | (xx.x) |

Note: Percent is based on the total number of patients in the Safety Population.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table1.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Completion date is date of death. Death reasons are recorded in categories stated.

Note to programmer: The number of patients who met all Inclusion/Exclusion criteria is based on response from page 12 of the CRF

Table 2

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

| Demographics | |
|-------------------------------------|------------|
| | N = xx (%) |
| Age at informed consent (yrs) | |
| N | XX |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | xx |
| Gender (%) | N |
| Female | xx (xx.x) |
| Male | xx (xx.x) |
| If Female: Child-bearing status (%) | N |
| Post-menopausal | xx (xx.x) |
| Surgically sterile | xx (xx.x) |
| Childbearing potential | xx (xx.x) |
| Unknown | xx (xx.x) |
| Race/ethnicity (%) | N |
| Black/Afro-Caribbean | xx (xx.x) |

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

| White/Caucasian Asian Other | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
|-----------------------------|-------------------------------------|
| Height (cm) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. | XX |
| Max. | xx |
| WHO performance status (%) | N |
| 0 | xx (xx.x) |
| 1 | xx (xx.x) |
| 2 | xx (xx.x) |
| 3 | xx (xx.x) |
| 4 | xx (xx.x) |

### **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Note: Percent is based on the number of patients who provided a response for each criteria.

Note: Age at informed consent derived using: Age (years) = integer part of ((patient informed consent date - date of birth + 1)/365.25). Full date of birth is used in the calculation, but only year of birth is listed.

Note: WHO performance status assessment

0=Asymptomatic, 1=Symptomatic but completely ambulatory, 2=Symptomatic <50% in bed during the day, 3=Symptomatic >50% in bed but not bedbound, 4=Bedbound.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table2.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 3a Melanoma Specific Medical History

| | N = XX (%) |
|--------------------------------------------------------------|------------|
| Time since initial diagnosis of current presentation (years) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | xx.x |
| Min. | xx |
| Max. | XX |
| Time since excision of primary lesion (years) | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | XX |
| Time since excision of sentinel node (years) | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | XX |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

| Max. | xx |
|---------------------------------------------------------------|----------|
| Time since resection of regional lymph node resection (years) | |
| N | xx |
| Mean | xx.x |
| SD | XX.XX |
| Median | XX.X |
| Min. | xx |
| Max. | xx |
| Stage of disease (%) | N |
| Stage III a | xx(xx.x) |
| Stage III b | xx(xx.x) |
| Stage III c | xx(xx.x) |
| Stage IV | xx(xx.x) |
| Unknown | xx(xx.x) |
| Other | xx(xx.x) |
| Primary lesion thickness (T type) (mm) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. | XX |
| Max. | XX |
| Presence of lymph node metastases (N type) (%) | N |
| Yes | xx(xx.x) |
| No | xx(xx.x) |
| Unknown | xx(xx.x) |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

| Current lesions (%) | N |
|-----------------------------------|----------|
| Yes | xx(xx.x) |
| No | xx(xx.x) |
| Unknown | |
| If Yes: Location of lesion(s) (%) | N |
| Location 1 | xx(xx.x) |
| Location 2 | xx(xx.x) |
| Location n | xx(xx.x) |

### **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Note: As patients may have more than one lesion in various locations they can be included in more than one location category.

Note: Percent is based on the number of patients who provided a response for each criteria.

Note: Time (years) since variables are calculated from Day 0 + 1 and divided by 365.25.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table3a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Locations listed under PELOC e.g. Lung.

Note to programmer: If stage is other and more information is provided include it in the other description or as a footnote.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

Note to programmer: Please add footnote if any 'time since' variables contain partial missing dates, see SAP section 8.2: Where day and month are not known for either date, calculation is based on year alone: Time since event (years) = (Year of Day 0 - Year of event) + 1/365.25, likewise if day is not known for either date, calculation is based on month and year only

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Table 3b

Significant Medical History since Completion of Study IMM-101-001

System Organ Class

| Preferred Term | N = xx (%) |
|---|---|
| Significant or clinically relevant medical history since completion of study IMM-101-001? | N |
| Yes | xx(xx.x) |
| No | xx(xx.x) |
| Unknown | xx(xx.x) |
| If Yes: | |
| System Organ Class | N |
| Preferred Term 1 | xx(xx.x) |
| Preferred Term 2 | xx(xx.x) |
| Preferred Term n | xx(xx.x) |

Note: Medical History is coded using MedDRA version xx.x.

Note: Percent is based on the number of patients in the Safety Population.

 $\label{lem:code:s:Services} Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table3b.sas \ ddmmmyy: hh:mm:ss \ ddmmmyy: hh:mm:sd \ ddmmmyy: hh:mm:s$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Please add relevant MedDRA version number in note to reflect version used at time of coding.

Note to programmer: Sort SOC and PT by decreasing incidence.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Table 4
Pre-study IMM-101 Administration Since Completion of Study IMM-101-001

| | N = xx (%) |
|---|---|
| Any IMM-101 administration(s) since the completion of the Phase 1 study IMM-101-001(%) Yes No | xx(xx.x)<br>xx(xx.x) |
| Number of patients who received at least 1 dose of: (%) | |
| xx.x mg | xx(xx.x) |
| xx.x mg | xx(xx.x) |
| xx.x mg | xx(xx.x) |
| Total number of doses administered over all patients at dose of: | |
| xx.x mg | XX |
| xx.x mg | XX |
| xx.x mg | XX |
| Total number of doses administered pre-study | xx |
| Total number of doses received per patient | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

| Median | XX.X |
|--------|------|
| Min. | XX |
| Max. | XX |

Note: Percent is based on the number of patients who provided a response for each criteria.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table4.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

### **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 5 Pre-Existing Injection Site Reaction(s)

| N=xx (%) |
|-----------|
| N |
| N |
| xx(xx.x) |
| xx(xx.x) |
| xx (xx.x) |
| N |
| xx(xx.x) |
| xx(xx.x) |
| xx(xx.x) |
| xx(xx.x) |
| xx (xx.x) |
| N |
| xx(xx.x) |
| xx(xx.x) |
| xx(xx.x) |

Note: Percent is based on the number of patients who provided a response for each criteria.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table5.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

#### Table 6

Summary of Anti-melanoma Cancer Therapies other than IMM-101 Whilst on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined) N=XX

| Number of patients with at least one other anti-cancer | v | (xx.x) |
|--------------------------------------------------------|---|--------|
| therapy | X | (XX.X) |
| Cancer Surgery | Х | (xx.x) |
| XXXX | X | (xx.x) |
| XXXX | X | (xx.x) |
| Chemotherapy | X | (xx.x) |
| XXXX | X | (xx.x) |
| Immunotherapy | X | (xx.x) |
| XXXX | X | (xx.x) |
| Radiotherapy | X | (xx.x) |
| XXXX | Х | (xx.x) |
| Radiofrequency Ablation | X | (xx.x) |

### **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

X = XX

Note: Anti-melanoma cancer Therapies include melanoma-related surgery, chemotherapy, radiotherapy, radiofrequency ablation and non-IMM-101 immunotherapy treatments ongoing or started on/after the first dose of IMM-101 in study IMM-101-001, including therapies during NPP (recorded as medical history since leaving study IMM-101-001) and during IMM-101-008.

Note: Therapies are counted once per therapy type per patient hence duplicates are not included in the table.

Note: Percent is based on the total number of patients in the Analysis Population.

XXXX

Note: MedDRA preferred terms are reported for procedures reported with AEs. Otherwise, verbatim terms are reported. Preferred Term is coded using MedDRA version 18.1

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table6.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxx.sas7bdat, S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxxx.sas7bdat,

S:\Services\Immodulon\IMM-101-008\DataManagement\DataEntry\Coding Files\cancer coding lookup xx xxx xxxx.sas7bdat,

Note to programmer: Please update data footnote with appropriate file directory. Please sort by decreasing incidence at therapy type and treatment level. Non-cancer treatments and immunotherapy IMM-101 will be excluded from this table.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Table 7
On-Study IMM-101 Administration

| | Visit 1 | Visit N |
|----------------------------|----------|----------|
| | N | N |
| IMM-101 dose administered? | | |
| No | xx(xx.x) | xx(xx.x) |
| Yes | xx(xx.x) | xx(xx.x) |
| If Yes: | | |
| Full dose (1 mg) | xx(xx.x) | xx(xx.x) |
| Reduced dose (<1 mg) | xx(xx.x) | xx(xx.x) |

Note: The percent will be based on the number of patients available at each visit who provide a response.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table7.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Where 'Visit N' appears add additional columns as required. If too many Visits for columns create sets of rows for each visit number.

### **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

# Table 8 Overall Survival

| Total number of patients | XX |
|-------------------------------|----------------------------|
| Number of deaths | XX |
| Number of censored events | xx |
| Median survival time (95% CI) | xx.x ( $xx.xx$ , $xx.xx$ ) |
| 25% survival time (95% CI) | xx.x (xx.xx, xx.xx) |
| 75% survival time (95% CI) | xx.x (xx.xx, xx.xx) |

Note: The summary statistics for survival time have been derived based on the Kaplan-Meier product limit survival estimates.

Note: Overall survival (years) is calculated as ((date of death or censored date) - Day 0 + 1)/365.25.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table8.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Table 9a

Analysis Population: Safety Population

| Exposure | |
|-------------------------------------------|--------|
| 2 111 1 | N = xx |
| Time on study (years) | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | xx |
| Overall study drug exposure (months) | |
| N | xx |
| Mean | XX.X |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | xx |
| Total no. IMM-101 doses received on study | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Median xx.x Min. xx Max. xx

Note: Time on study (years) = (date of completion (i.e. death on study)/date of withdrawal - Day 0 + 1)/365.25.

Overall Exposure (months) = (date of last dose - date of first dose in study IMM-101-008 + 1)/30.4375.

Total number of doses received = sum of the doses (full or part doses counted as 1 dose) received, as reported in the CRF.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table9a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

Table 9b

Time on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined)

Overall study drug exposure (months)

 N
 X

 Mean
 xx.xx

 StD
 xx.xxx

 Median
 xx.xx

 Min.
 xx.x

 Max.
 xx.x

Note: Overall study drug exposure is derived as follows:

Overall study drug exposure (months) = (date of last dose in study IMM-101-008 - date of first dose in study IMM-101-001 + 1)/30.4375.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\ Table9b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxx.sas7bdat,

S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxx.sas7bdat,

S:\Services\Immodulon\IMM-101-008\SDTM\ xxxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Table 10a
Summary of Treatment Emergent Adverse Events

| | N = xx (%) |
|---|---|
| Number of patients with treatment emergent adverse events (%) | xx(xx.x) |
| Number of treatment emergent adverse events | XX |
| Number of patients with treatment emergent adverse events related to the study drug (%) | xx(xx.x) |
| Number of treatment emergent adverse events related to the study drug | XX |
| Number of patients with serious treatment emergent adverse events (%) | xx(xx.x) |
| Number of serious treatment emergent adverse events | XX |
| Number of patients with serious treatment emergent adverse events relating to the study drug (%) | xx(xx.x) |
| Number of serious treatment emergent adverse events relating to the study drug | XX |
| Number of patients with treatment emergent adverse events leading to withdrawal or death (%) | xx(xx.x) |
| Number of treatment emergent adverse events leading to withdrawal or death | XX |
| Number of patients with treatment emergent adverse events of NCI CTCAE $\geq$ Grade 3 (%) | xx(xx.x) |
| Number of treatment emergent adverse events of NCI CTCAE ≥ Grade 3 | XX |

Note: Treatment emergent AEs are all those reported during the study. Related AEs are defined as events that are definitely, probably or possibly related to study drug or with an unknown relationship.

Note: CTCAE - Common Toxicity Criteria for Adverse Events CTCAE decode.

Note: Percent is based on total number of patients in the Safety Population.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10b Treatment Emergent Adverse Events

| System Organ Class/ | |
|---------------------------------------------------------------|-----------|
| Preferred Term | N = XX |
| | n(%) m |
| Number of patients with treatment emergent adverse events (%) | xx(xx.x) |
| Total Number of treatment emergent adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

#### Table 10c

Treatment Emergent Adverse Events with NCI CTCAE Grade ≥ 3

| System Organ Class/ Preferred Term | N = xx<br>n(%) m |
|---|---|
| Number of patients with treatment emergent adverse events of NCI CTCAE $\geq$ Grade 3 Total Number of treatment emergent adverse events of NCI CTCAE $\geq$ Grade 3 | xx (xx.x)<br>xx |
| System Organ Class Preferred Term | n(xx.x) m<br>n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

Note: Common Toxicity Criteria for Adverse Events CTCAE decode. 1. Mild, 2. Moderate, 3, Severe, 4. Life Threatening, 5. Death

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10c.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10d Treatment Emergent Adverse Events Related to IMM-101

| System Organ Class/ | N = XX |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with treatment emergent, related adverse events (%) | xx(xx.x) |
| Total Number of treatment emergent, related adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study. Related AEs are defined as events that are definitely, probably or possibly related to study drug or with an unknown relationship.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10d.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10e Treatment Emergent Serious Adverse Events

| System Organ Class/ | N = xx |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with serious, treatment emergent adverse events (%) | xx(xx.x) |
| Total Number of serious, treatment emergent adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

 $\label{thm:ss} \textbf{Code: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash Analysis\backslash Development\backslash Code\backslash Table 10e.sas \ ddmmmyy: hh:mm:ss} \\$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

#### Table 10f

Treatment Emergent Adverse Events Leading to Withdrawal or Death

| System Organ Class/ | N = XX |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with treatment emergent adverse events leading to withdrawal or death (%) | xx(xx.x) |
| Total Number of treatment emergent adverse events leading to withdrawal or death | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; <math>m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10f.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10g Treatment Emergent Non-serious Adverse Events

| System Organ Class/ | |
|---|---|
| Preferred Term | N = XX |
| | n(%) m |
| Number of patients with treatment emergent non-serious adverse events (%) | xx(xx.x) |
| Total Number of treatment emergent non-serious adverse events | XX |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with a non-serious AE; <math>m = number of non-serious AEs.

Hence if a patient has multiple non-serious AEs only one occurrence per person will contribute to 'n', but all occurrences will

be counted under  $\mbox{'m'}$  as this is the total number of non-serious events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent non-serious AEs are all those reported during the study.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10g.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

Note to programmer: Please add relevant version number in MedDRA note to reflect version used at time of coding

Note to programmer: All non-serious AEs are to be excluded from this summary table.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

#### Table 10h

Treatment-related Treatment Emergent Adverse Events (IMM-101-001 and IMM-101-008 Combined)

| System Organ Class/ | N = xx |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with treatment-related treatment emergent adverse events (%) | xx(xx.x) |
| Total Number of treatment-related treatment emergent adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version 18.1.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported at/after first IMM-101 dosing in study IMM-101-001. Related AEs are defined as AEs that are definitely, probably or possibly related to study drug or with an unknown relationship.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\ Table10h.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Data: S:\Services\Immodulon\IMM-101-001\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory. Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

Table 11
On-Study Injection Site Reaction(s)

| | Visit 1<br>N = xx (%) | Visit 2<br>N = xx (%) | Visit N<br>N = xx (%) |
|---|---|---|---|
| Is the injection site reaction from previous IMM-101 dose(s) visible? | N | N | N |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| If visible, are daily activities affected? | N | N | N |
| Not at all | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderately | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Quite badly | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intolerably | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Worsening with repeated doses of IMM-101? | N | N | N |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Sure | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Wound care required? | N | N | N |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Percent are based on the number of patients available at each visit who provided a response.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table11.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Where 'Visit N' appears add additional columns as required, or reverse rows and columns if visits large in number, so rows become visits and variables are in the columns.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

# Listing 1 Patient Disposition

| Unique<br>Patient ID | Consent Date<br>(DD-MM-<br>YYYYTHH:MM) | Versio<br>n<br>Number | Off-Study<br>Date<br>(DD-MM-YYYY) | Off-<br>Study<br>Status | Time on<br>Study<br>(years) | Overall<br>Study<br>drug<br>exposure<br>(months) | Total no. IMM- 101 Doses receiv ed on Study | Reason<br>for<br>Completio<br>n (death)<br>or<br>Withdrawa | All adverse events<br>followed for at<br>least 30 days<br>after study<br>completion/withdra<br>wal | Principal Investiga tor Sign off Date (DD-MM- YYYY) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | xxxxx | XX | XX | XX | xxxxx | xxxxx | DD-MM-<br>YYYY |
| XXXXX | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | XXXXX | XX | XX | XX | XXXXX | xxxxx | DD-MM-<br>YYYY |
| XXXXX | DD-MM-YYYY HH:MM | xx | DD-MM-YYYY | XXXXX | XX | XX | XX | XXXXX | xxxxx | DD-MM-<br>YYYY |
| XXXXX | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | XXXXX | XX | XX | XX | XXXXX | xxxxx | DD-MM-<br>YYYY |
| xxxxx | DD-MM-YYYY HH:MM | xx | DD-MM-YYYY | XXXXX | xx | xx | xx | xxxxx | xxxxx | DD-MM- |
| xxxxx | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | XXXXX | XX | XX | XX | xxxxx | xxxxx | YYYY<br>DD-MM-<br>YYYY |

Note: Time on study (years) = (date of completion (i.e. death on study)/date of withdrawal - Day 0 + 1)/365.25.

Overall Exposure (months) = (date of last dose - date of first dose in study IMM-101-008 + 1)/30.4375.

Total number of doses received = sum of the doses (full or part doses counted as 1 dose) received, as reported in the CRF.

Note: The trial was terminated in Dec-2018 as no further meaningful data was being collected nor was likely to be collected in the future.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing1.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Off-Study Status should be either 'Completed Study - patient died' or 'Withdrew'.

Note to Programmer: Where applicable, separate date from time using a space.

Note to Programmer: Status at completion/withdrawal: If reason is AE/unacceptable toxicity, Investigator decision or Patient did not meet INC/EXC criteria, please include specify text. If reason is other please include reason/description where applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 2
Demographics

| Unique<br>Patient<br>ID | Year of<br>Birth<br>(YYYY) | Age at Informed Consent (years) | Race/<br>Ethnicity | Gender | Child-<br>bearing<br>Status | Height<br>(cm) | WHO<br>Performance<br>Status |
|---|---|---|---|---|---|---|---|
| ' | | | | | | | |
| XXXXX | YYYY | XX | XXXXX | XXXXX | XXX | XXX | X |
| XXXXX | YYYY | XX | XXXXX | XXXXX | XXX | XXX | X |

Note: Age at informed consent will be derived using; Age (years) = integer part of ((patient informed consent date - date of birth + 1)/365.25).Note: Full date of birth is used in the calculation, but only year of birth is listed.

Note: WHO performance status assessment

0=Asymptomatic, 1=Symptomatic but completely ambulatory, 2=Symptomatic <50% in bed during the day, 3=Symptomatic >50% in bed but not bedbound, 4=Bedbound.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing2.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: If Race/ethnicity was recorded as 'Other' on the CRF then the response provided should be listed.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Not Applicable

# Listing 3a Inclusion/Exclusion Questions

| Question<br>Number | Inclusion/<br>Exclusion<br>Criteria | Question |
|---|---|---|
| 1 | Inclusion | Were previously enrolled in Study IMM-101-001. |
| 2 | Inclusion | Give consent to make their disease and treatment history for the intervening period between their completion of Study IMM-101-001 and enrolment in this study available to the Sponsor. |
| 3 | Inclusion | Give signed informed consent for participation in the study. |
| 1 | Exclusion | Female patient of child-bearing potential who is not, in the opinion of the Investigator, using an approved method of birth control (e.g., physical barrier [patient and partner], contraceptive pill or patch, spermicide and barrier, or intrauterine device [IUD]). Those patients that utilise hormonal contraceptives must have used the same method for at least three months before additional barrier contraception (as described above) is discontinued from being used concomitantly with the hormonal contraception. Patient of non-child-bearing potential are defined as having 12 month amenorrhoea or are surgically sterile. |
| 2 | Exclusion | Female patient who is pregnant, breast feeding or planning a pregnancy during the course of the study. A pre-treatment urine pregnancy test measuring human chorionic gonadotrophin (HCG) must be negative. |
| 3 | Exclusion | Patient is unable or unwilling to comply with the protocol. |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing3a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Listing 3b
Inclusion/Exclusion Criteria

| Unique<br>Patient ID | Date of<br>Collection<br>(DD-MM-YYYY) | Question<br>Number | Inclusion/<br>Exclusion<br>Criteria | Criteria<br>Met?<br>(Y/N) |
|---|---|---|---|---|
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| xxxxx | DD-MM-YYYY | XX | xxxxx | XX |

Note: Reference Listing 3a for Inclusion/Exclusion Criteria Questions

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing3b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Inclusion / Exclusion criteria will be used to identify which questions are inclusion criteria and which are exclusion criteria. Only numbers should listed in the question number column.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 3c Inclusion/Exclusion Criteria Confirmation

| Unique<br>Patient<br>ID | Eligibility<br>confirmation | Eligibility<br>Confirmation<br>Date(DD-MM-<br>YYYY) | Eligibility<br>Re-confirmation | Eligibility<br>Re-confirmation<br>Date(DD-MM-YYYY) |
|---|---|---|---|---|
| xxxxx | xxxxx | DD-MM-YYYY | XXXXX | DD-MM-YYYY |
| XXXXX | XXXXX | DD-MM-YYYY | XXXXX | DD-MM-YYYY |
| XXXXX | XXXXX | DD-MM-YYYY | xxxxx | DD-MM-YYYY |

 ${\tt Code: S:\Services\setminus Immodulon\setminus IMM-101-008\setminus Analysis\setminus Development\setminus Code\setminus Listing 3c.sas \ ddmmmyy:hh:mm:ss.}$ 

 ${\tt Data: S:\Services\setminusImmodulon\setminusIMM-101-008\setminus xxxxx.sas7bdat}$ 

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Eligibility re-confirmation date is date of Day 0 (CRF page 11)

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

## Listing 4ai Melanoma Specific Medical History

| Unique<br>Patient<br>ID | Date of Initial Diagnosis of Current Presentation (DD-MM-YYYY) | Date of Excision of Primary Lesion (DD-MM-YYYY) | Date of Excision of Sentinel Node (DD-MM-YYYY) | Date of<br>Regional Lymph<br>Node Resection<br>(DD-MM-YYYY) | Date of Last<br>CT Scan<br>(DD-MM-YYYY) | Stage of<br>Disease | Primary<br>Lesion<br>Thickness<br>(T type) | Presence of<br>Lymph Node<br>Metastases<br>(N Type) |
|---|---|---|---|---|---|---|---|---|
| xxxxx | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | xxxxx | xxxxx | xxxxx |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | XXXXX |

Note: Dates have been listed where provided.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing4ai.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown/Not resected/Not excised/other specified text should be presented in the appropriate columns where applicable.

Note to programmer: Date of last CT scan is from CRF page 4: Disease and Treatment History

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

# Listing 4aii Melanoma Specific Medical History Continued

| | Ti | me (years) | since | | Lesion(s) details | | | | 3 |
|---|---|---|---|---|---|---|---|---|---|
| Unique | Initial | Excision | Excision | Regional | Presence | Melanoma | Longest | Shortest | Location |
| Patient | Diagnosis of | of | of | Lymph | of Current | Lesion | Diameter | Diameter | of Lesion |
| ID | Current | Primary | Sentinel | Node | Lesions | Number | (mm) | (mm) | |
| | Presentation | Lesion | Node | Resection | | | | | |
| XXXXX | XX | XX | XX | XX | XXXXX | 1 | X.XX | X.XX | XXXXX |
| | | | | | | 2 | X.XX | X.XX | XXXXX |
| | | | | | | 3 | X.XX | X.XX | XXXXX |
| | | | | | | 4 | X.XX | X.XX | XXXXX |
| XXXXX | XX | XX | XX | XX | XXXXX | 1 | X.XX | X.XX | XXXXX |
| | | | | | | 2 | X.XX | X.XX | XXXXX |

Note: Time (years) since variables are calculated from Day 0 + 1 and divided by 365.25.

Note: The screening assessment visible cutaneous lesions measurements were not recorded. Post screening assessment of lesions was not requested in the CRF.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing4aii.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Please add footnote if any 'time since' variables contain partial missing dates, see SAP section 8.2: Where day and month are not known for either date, calculation is based on year alone: Time since event (years) = (Year of Day 0 - Year of event) + 1/365.25.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Listing 4b
Significant Medical History since Completion of Study IMM-101-001

| Unique<br>Patient<br>ID | No<br>Significant<br>Medical<br>History | Body<br>system<br>Code* | Diagnosis | Preferred<br>Term | System<br>Organ<br>Class | Treatment | Start Date<br>(DD-MM-<br>YYYY) | Stop Date<br>(DD-MM-YYYY) | Anti-melanoma<br>Cancer Therapy |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | xxxxx | XXXXX | xxxxx | xxxxx | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |

Note: \*As recorded by the investigator

Note: Significant medical history includes all relevant anti-melanoma cancer therapy (radiotherapy, cancer surgery, chemotherapy, immunotherapy etc.) other than IMM-101 since finishing study IMM-101-001. Anti-melanoma cancer therapies are determined by the Sponsor's medical reviewer and flagged in the Anti-melanoma Cancer Therapy column.

Note: Preferred terms are coded using MedDRA version xx.x

Note: Ongoing is recorded as free text in the CRF where provided.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing4b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown should be presented in the appropriate date columns were applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

Listing 5
Pre-Existing Injection Site Reaction(s) Assessed at Screening

| Unique<br>Patient<br>ID | Injection Site<br>Reaction Present | Counts Right<br>Deltoid | Counts Left<br>Deltoid | Do(es) The Local<br>Reaction(s) Affect<br>Daily Activities? | Comments<br>(where<br>applicable) |
|---|---|---|---|---|---|
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |

Note: Counts = Number of pre-existing injection site reactions present.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing5.sas ddmmmyy:hh:mm:ss

 ${\tt Data: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash xxxxx.sas7bdat}$ 

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Listing 6
Screening Urine Pregnancy Test Results

| _ | Unique Patient ID | Result | Reason Test Not<br>Performed (if<br>applicable) |
|---|---|---|---|
| | xxxxx | XXXXX | xxxxx |
| | xxxxx | xxxxx | XXXXX |
| | xxxxx | XXXXX | XXXXX |
| | xxxxx | XXXXX | xxxxx |
| | xxxxx | xxxxx | XXXXX |
| | xxxxx | xxxxx | xxxxx |
| | xxxxx | xxxxx | ××××× |
| | AAAXX | AAAAX | AAXXX |
| | XXXXX | XXXXX | XXXXX |

Note: Test performed should be one of Yes, No, Not done or N/A (where N/A represents either males, or females who have had a hysterectomy)

 ${\tt Code: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash Analysis\backslash Development\backslash Code\backslash Listing 6.sas \ ddmmmyy:hh:mm:ss}$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Reason test not preformed is recorded in LBREASND.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y Analysis Population: Safety Population

> Listing 7 Disease and Treatment History at Screening

| Unique<br>Patient ID | Any medication within last 28 days ongoing or ceased? | Any IMM-101 administrations since patient completed Phase 1 study IMM-101- 001? | Significant or clinically relevant medical history since completing IMM-101-001? | History of severe local reaction following previous administrations of IMM-101? | Comments | Date of last CT scan<br>(DD-MM-YYYY) |
|---|---|---|---|---|---|---|
| XXXXX | XX | XX | xxxxx | XXXXX | XXXXX | DD-MM-YYYY |
| XXXXX | XX | XX | xxxxx | xxxxx | XXXXX | DD-MM-YYYY |
| XXXXX | XX | XX | xxxxx | xxxxx | XXXXX | DD-MM-YYYY |
| XXXXX | XX | XX | XXXXX | xxxxx | XXXXX | DD-MM-YYYY |
| xxxxx | XX | XX | XXXXX | xxxxx | xxxxx | DD-MM-YYYY |
| xxxxx | XX | XX | XXXXX | xxxxx | xxxxx | DD-MM-YYYY |
| xxxxx | XX | XX | XXXXX | xxxxx | xxxxx | DD-MM-YYYY |
| xxxxx | XX | XX | xxxxx | xxxxx | xxxxx | DD-MM-YYYY |

Note: Refer to Listing 4b for CRF page 7 comments.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing7.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: If unknown is recorded, for date of last CT scan, it should be included in the column were applicable.

Note to programmer: Date of last CT scan is from CRF page 8: Melanoma Specific History.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Listing 8a Previous Medications

| Unique<br>Patient ID | Previous<br>Medications<br>Taken is None | Reported<br>Name of Drug | Dose | Dose<br>Units | Indication | Start<br>Date<br>(DD-MM-<br>YYYY) | End Date<br>(DD-MM-<br>YYYY) | Was the<br>Mediation Taken<br>and Stopped<br>Before 14 days<br>Prior to Day 0? | Anti-melanoma<br>Cancer Therapy |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | x | xxxxx | | | xxxxx | DD-MM- | DD-MM- | X | |
| | | | X.XX | XX | | YYYY | YYYY | | |
| XXXXX | X | XXXXX | X.XX | | XXXXX | DD-MM- | DD-MM- | X | XXXXXXX |
| | | | | XX | | YYYY | YYYY | | |
| XXXXX | X | XXXXX | X.XX | | XXXXX | DD-MM- | DD-MM- | X | |
| | | | | XX | | YYYY | YYYY | | |

Note: Previous medications are all medications (prescription/non-prescription), including vitamins, drugs of abuse, and dietary supplements taken and stopped within 14 days prior to the end of screening procedures (i.e. Day 0). Any previous medications taken and stopped before 14 days prior to Day 0 have been flagged and included in the listing.

Note: Anti-melanoma cancer therapies are determined by the Sponsor's medical reviewer and flagged in the Anti-melanoma Cancer Therapy column.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing8a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown should be presented in the appropriate date columns were applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

## Listing 8b Concomitant Therapies

| Unique<br>Patient<br>ID | Reported Name<br>of Drug | Indication | Dose | Dose<br>Units | Dosing<br>Frequency | Start Date<br>(DD-MM-YYYY) | End Date<br>(DD-MM-YYYY) | Anti-melanoma<br>Cancer Therapy |
|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxxx | XXXXX | x.xx | XX | xxxxx | DD-MM-YYYY | DD-MM-YYYY | XXXXXXX |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXXXXX |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |

Note: Concomitant Medications are all medications (prescription/non-prescription), including vitamins, and dietary supplements and surgical procedures ongoing or started on/after Day 0.

Note: Anti-melanoma cancer therapies are determined by the Sponsor's medical reviewer and flagged in the Anti-melanoma Cancer Therapy column.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing8b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown should be presented in the appropriate date columns were applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 9
Previous IMM-101 Administrations Since Completion of Study IMM-101-001

| Unique Patient<br>ID | Date of Last Administration of IMM-101 in Study IMM-101-001 (DD-MM-YYYY) | Administration Date of IMM-101 Since Completion of IMM-101-001 (DD-MM-YYYY) | Dose<br>(mg) | Injection<br>Site (R or<br>L Deltoid) |
|---|---|---|---|---|
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | X.XX | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | x.xx | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | X.XX | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | x.xx | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | X.XX | xxxxx |

Note: IMM-101 administrations since completion of IMM-101-001 were taken whilst patient was in Named Patient Programme and injection location was not recorded during this period.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing9.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: If date of administration is recorded as not known, present Unknown in place of date for the relevant dose.

Note to programmer: Date of last administration of IMM-101 in IMM-101-001 study should be displayed only once per patient.

S:\Services\Immodulon\IMM-101-008\SMF\SAP\IMM-101-008\_ SAPvFinal 1.1


## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

# Listing 10 On-Study IMM-101 Administration

| Unique<br>Patient<br>ID | Visit<br>Name/<br>Number | Visit Date | Date of Last<br>Dose of IMM-<br>101<br>(DD-MM-YYYY) | Have at Least 14 Days Passed Since Last Dose? | Time Elapsed Between This and Previous Dose (days) | Dose<br>Administered<br>(Y/N) | Dose<br>(mg) | Dose<br>Changed<br>From<br>Previous<br>Dose | Reason for<br>Dose<br>Reduction or<br>Delay (if<br>applicable) | Injection<br>Site |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | xx | x.xx | Х | xxxxx | xxxxx |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | x.xx | Х | xxxxx | xxxxx |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | Х | xxxxx | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | XXXXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | Х | XXXXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | XXXXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | xxxxx | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | xxxxx | XXXXX |

Note: Time elapsed since previous dose (days) = (date of current dose - date of previous dose + 1).

Note: Dose changed from previous dose; I = increased, D = decreased (when compared with previous IMM-101 dose).

Note: Reasons for dose increases were also recorded in the CRF, as indicated.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing10.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Injection site should include right/left deltoid and upper/lower.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 11 On-Study Disease Assessment

| Unique<br>Patient ID | Visit<br>Name/Number | Visit Date<br>(DD-MM-YYYY) | Has a CT Scan been conducted since the last visit? (Y/N) | If yes, at the investigator's discretion, please indicate disease status compared to the last assessment | Comment (if applicable) |
|---|---|---|---|---|---|
| xxxxx | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | XXXXX | xxxxx |
| XXXXX | XXXXX | DD-MM-YYYY | xx | xxxxx | xxxxx |

Note: Per protocol Investigator was asked to assess the presence of metastatic disease (if applicable) periodically following CT or MRI scan performed as routine standard of care.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing11.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

## Listing 12 Adverse Events

| AE<br>No. | Reported<br>AE term | Preferred<br>Term | System<br>Organ<br>Class | Intensity<br>(CTCAE) | Seriousness<br>(N/Y) | Reason for<br>Seriousness/<br>Details if<br>other | Relationship<br>to Study<br>Drug | Start Date/Time<br>(DD-MM-YYYY<br>HH:MM) | End Date/Time (DD-MM-YYYY HH:MM) | Outco<br>me | Sequelae |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | xxxxx | xxxxx | xxxxx | xxxxx | XX | xxxxx | xxxxx | DD-MM-YYYY HH:MM | DD-MM-YYYY HH:MM | xxxxx | xxxxx |
| XX | XXXXX | XXXXX | xxxxx | XXXXX | XX | XXXXX | XXXXX | DD-MM-YYYY HH:MM | DD-MM-YYYY HH:MM | XXXXX | xxxxx |
| XX | XXXXX | XXXXX | XXXXX | XXXXX | XX | XXXXX | XXXXX | DD-MM-YYYY HH:MM | DD-MM-YYYY HH:MM | XXXXX | XXXXX |
| | No. xx xx xx xx xx xx xx | XX XXXXX XX XXXXX | No. AE term Term xx xxxxx xxxxx xx xxxxx xxxxx | No. AE term Term Organ Class xx xxxxx xxxxx xxxxx xx xxxxx xxxxx xxxxx | No. AE term Term Organ (CTCAE) xx xxxxx xxxxx xxxxx xx xxxxx xxxxx xxxxx | No. AE term Term Organ Class (CTCAE) (N/Y) xx xxxxx xxxxx xxxxx xxxxx xxxxx xx xx xxxxx xxxxx xxxxx xx xx xx xxxxx xxxxx xxxxx xx xx xxxxx xxxxx xx | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ Details if other xx xxxxx xxxxx xxxxx xxxxx xxxxx xx xxxxx xxxxx xxxxx xxxxx | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ other to Study Drug other xx xxxxx xxxxxx xxxxxx xxxxxx xxxxxx | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ other to Study (DD-MM-YYYY HH:MM) xx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ betails if other to Study (DD-MM-YYYY (DD-MM-YYYY HH:MM) (DD-MM-YYYY HH:MM) HH:MM) xx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM DD-MM-YYYY HH:MM | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ to Study Drug HH:MM) HH:MM) xx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx xxxx |

Note: Treatment emergent AEs are all those reported during the study. Sequelae column also contains comments recorded in the sequelae field of the CRF.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Common Toxicity Criteria for Adverse Events CTCAE code. 1. Mild, 2. Moderate, 3. Severe, 4. Life Threatening, 5. Death

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing12.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Where applicable, separate date from time using a space.

Note to Programmer: If Reason for seriousness is other please include reason/description.

Note to Programmer: Intensity should be occupied with text, the numeric CTCAE codes are provided in a note.

Note to programmer: Please add relevant version number in MedDRA note to reflect version used at time of coding.

Note to programmer: If necessary, break table over two pages with each new section of the table displaying Unique Patient ID, AE No., Reported AE term, Treatment Emergent, Preferred Term and System Organ Class.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Listing 13 On-Study Injection Site Reaction(s)

| Unique<br>Patient<br>ID | Visit<br>Name/<br>Number | Visit Date<br>(DD-MM-YYYY) | Date Last Dose of IMM-101 Administered (DD-MM-YYYY) | Is/are Injection Site Reaction(s) Visible From Previous Doses(s) of IMM-101? | Do(es) the Local Reaction(s) Affect Daily Activities? | Are Injection Site<br>Reactions Becoming<br>More Troublesome<br>With Repeated<br>Doses of IMM-101 | Wound Care<br>Required | Description<br>of Wound<br>Care<br>Provided |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | XXXXX | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | xxxxx | XXXXX | XXXXX | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | xxxxx | XXXXX | xxxxx | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | xxxxx | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | XXXXX | XXX | xxxxx |

 ${\tt Code: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash Analysis\backslash Development\backslash Code\backslash Listing 13.sas \ ddmmmyy: hh:mm:ss} \\$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Listing 14
Concomitant Medication and Adverse Event Checks

| Unique<br>Patient ID | Visit<br>Name/Number | Visit<br>Date<br>(DD-MM-YYYY) | Any medication (prescription or non-prescription) started or ceased since the last dose of IMM-101? (Y/N/Unknown) | Other than a local reaction, did the patient have any concurrent sign(s), symptoms(s), and or disease(s)? (Y/N) |
|---|---|---|---|---|
| xxxxx | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |

Note: UK, U = Unknown.

 ${\tt Code: S:\Services\setminus Immodulon\setminus IMM-101-008\setminus Analysis\setminus Development\setminus Code\setminus Listing 14.sas \ ddmmmyy: hh:mm:ss} \\$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Listing 15 Study Visits and Visit Checklists

| Unique Patient<br>ID | Visit<br>Name/Number | Visit Date (DD-MM-YYYY) | Number of weeks<br>elapsed since last<br>visit (where<br>applicable) | Checklist Item | Completed (Y/N) |
|---|---|---|---|---|---|
| xxxxx | xxxxx | DD-MM-YYYY | XX | xxxxx | XX |
| xxxxx | xxxxx | DD-MM-YYYY | XX | xxxxx | XX |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing15.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Include Date of Consent for patient transfer to Site 2, date of first visit at Site 2 and nominal visit number according to CRF entries, in chronological order in the listing (see Immodulon file note FN47).

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

Note to programmer: All visits should be listed. Checklist items text to be stated in full. If text too long, add a key on separate listing 15a or similar.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 16
Blood Sample for Immunological Markers

| Unique Patient ID | Visit Name/<br>Number | Visit Date<br>(DD-MM-YYYY) | Blood Sample Taken?<br>(Y/N) | Volume (mL) |
|---|---|---|---|---|
| xxxxx | XXXXX | DD-MM-YYYY | XX | XX.X |
| XXXXX | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| XXXXX | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing16.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

# Listing 17 Post-Study Long Term Survival Status

| Unique Patient<br>ID | Date of Consent For<br>Data Collection | Date of Assessment<br>of Status<br>(DD-MM-YYYY) | Survival Status | If Death, Date of Death (DD-MM-YYYY) | If Death,<br>Cause of<br>Death | Investigator<br>Signature<br>Date<br>(DD-MM-YYYY) |
|---|---|---|---|---|---|---|
| xxxxx | XXXXX | DD-MM-YYYY | xxxx | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | xxxx | DD-MM-YYYY | XXXXX | XXXXX |

 $\label{lem:code:s:Services} Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing17.sas \ ddmmmyy:hh:mm:ss$ 

 ${\tt Data: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash xxxxx.sas7bdat}$ 

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Data is recorded on Post-study Survival Status CRF, with multiple rows per patient (depending on number of occasions long term survival status is assessed).

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 18
Additional Comments Recorded

| Unique Patient<br>ID | Related Domain | Visit at which comment recorded | Date of Visit<br>(DD-MM-YYYY) | Associated Variable | Comment |
|---|---|---|---|---|---|
| xxxxx | XXXX | xxxxx | DD-MM-YYYY | xxxx | XXXXX |
| XXXXX | xxxx | XXXXX | DD-MM-YYYY | XXXX | XXXXX |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing18.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Data is recorded as free text comments on the CRF.

Note to programmer: Please sort the listing by patient ID and related domain.

Note to programmer: For any comment relating to AEs, please put the 'AE xx:' in front of the comment.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y Analysis Population: Safety Population

Figure 1a Panel Plot of On-Study IMM-101 Doses by Patient



Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Figure1a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: A plot for each patient should be produced (with patient number in the subtitle for each plot) and all plots should be displayed in a panel plot (2x5). Each dose should be marked on the line plot by an 'X' or similar.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y Analysis Population: Safety Population

Figure 1b All IMM-101 Dosing Administrations (IMM-101-001 and IMM-101-008 Combined)



Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\ Figure1b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\ xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: A plot for each patient should be produced (with patient number in the subtitle for each plot) and all plots should be displayed in a panel plot (2x5 landscape format). Each dose should be marked on the line plot by an 'X' or similar. Standard axes should be used across the plots.
## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Figure 2
Kaplan Meier Curve of Overall Survival



Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Figure2.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Add Label along X-axis: Time (Years) after Day 0 date (X-axis range according to the time to event). Add Y-axis Proportion Alive. Include markers for withdrawn/censored patients.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

**Customer:** Immodulon Therapeutics Limited **Information Type:** Statistical Analysis Plan

| Title: | Statistical Analysis Plan for IMM-101-008 (long-term follow-up [LTF] study) |
|---|---|
| Version | Amendment 1 |
| Effective Date: | 10 April 2019 |

**Description:** An open label long-term follow-up study of patients with melanoma who were previously enrolled in the Phase I study IMM-101-001 (first-in-human [FIH] study).

Author's Name, Title and Functional Area: Sarah Taggart, Statistician, Exploristics Ltd

Helen Amine-Eddine, Consultant Statistician, KataCliniKa Ltd

Moira Murphy, Statistician, Exploristics Ltd

Approved by:

Helen Amine-Eddine

Consultant Statistician, KataCliniKa Ltd on behalf of Immodulon Therapeutics Ltd

Helen Amine-Eddine

Ma- Ma. A

Moira Murphy

Statistician Exploristics Ltd 10 April 2019

\_\_\_\_

10 Apr2019

Date

Copyright 2019 Exploristics Limited. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

| Audit Trail For This Document | | | |
|---|---|---|---|
| Compiled by/Affiliation | Type of Change | Date | Version |
| Sarah Taggart | Creation | 06 January 2015 | 0.1 |
| Anne-Marie Duggan | Internal review | 18 February 2015 | 1.0 |
| Immodulon | Review | 28 April 2015 | 1.1 |
| Sarah Taggart | Updates based on clients' comments | 08 May 2015 | 2.0 |
| Sarah Taggart | Updates based on client TC (18 MAY 2015) | 28 May 2015 | 3.0 |
| Immodulon | Review | 12 June 2015 | 3.1 |
| Sarah Taggart | Updates based on client review and correspondence | 26 June 2015 | 3.2 |
| Anne-Marie Duggan | Internal review | 01 July 2015 | 3.3 |
| Sarah Taggart | Pre-Final Draft | 09 July 2015 | Pre-Final Draft |
| Immodulon | Review | 16 September<br>2015 | Final Draft 1 |
| Sarah Taggart | Updates following client review | 30 September<br>2015 | Final Draft 2 |
| Anne-Marie | Final internal review | 06 October 2015 | Final Review |
| Sarah Taggart | Updates following final review | 07 October 2015 | Final |
| Effective Date | | 08 October 2015 | Final |
| Immodulon | Updates following review of SAP prior to final database lock and including relevant tables including IMM-101-001 and IMM-101-008 data for the Safety population of IMM-101-008 study, from the retired SAP Addendum. | 28 January 2019 | Amendment 1,<br>Draft 1 |
| Exploristics Ltd | Review | 11 February 2019 | Amendment 1,<br>Draft 1 |
| Immodulon | Incorporation of clarifications received following Exploristics review and Immodulon review comments | 11 February 2019 | Amendment 1,<br>Draft 2 |
| Exploristics Ltd | Final internal review | 14 March 2019 | Amendment 1,<br>Draft 3 |
| Clare Gleeson | Review (incorporating review by Exploristics Ltd) | 14 March 2019 | Final Draft |
| Effective Date | Incorporation of review comments and approval | 10 April 2019 | Final Amendment 1 |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

## **Table of Contents**

| ABBREVIATIONS | 4 |
|--------------------------------------------------------------|----|
| 1. INTRODUCTION | 5 |
| 2. STUDY OBJECTIVE(S) AND ENDPOINT(S) | 6 |
| 2.1 Study Objective(s) | 6 |
| 2.2 Study Endpoint(s) | 6 |
| 3. STUDY DESIGN | 7 |
| 4. PLANNED ANALYSES | 7 |
| 5. SAMPLE SIZE CONSIDERATIONS | 8 |
| 6. ANALYSIS POPULATIONS | 8 |
| 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES | 8 |
| 8. DATA HANDLING CONVENTIONS | 9 |
| 8.1 Premature Withdrawal and Missing Data | 9 |
| 8.3 Derived and Transformed Data | 10 |
| 9. DESCRIPTIVE STATISTICS | 13 |
| 9.1 Disposition of Patients | 13 |
| 9.2 Demographic and Baseline Characteristics | 13 |
| 9.3 Study Treatment, Exposure and Safety Outputs | 13 |
| 10. ANALYSIS CORRESPONDING TO THE STUDY OBJECTIVES | 15 |
| 11. PROTOCOL DEVIATIONS AND DEVIATIONS FROM PLANNED ANALYSIS | 16 |
| 12. REFERENCES | 16 |
| 13. ATTACHMENTS | 17 |
| 13.1 Table of Contents for Data Display Specifications | 17 |
| 13.2 Data Display Specification | 19 |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

## **ABBREVIATIONS**

| ADaM | Analysis Data Model |
|---------|------------------------------------------------------------|
| | Analysis Data Model |
| AE | Adverse Event |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| FIH | First-in-human |
| LTF | Long-term follow-up |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| NCI | National Cancer Institute |
| NPP | Named Patient Programme |
| OS | Overall Survival |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| TFL | Tables, Figures and Listings |
| Yrs | Years |

Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

#### 1. INTRODUCTION

The study explores the long-term safety and tolerability of continued administration of IMM-101 in patients who were previously enrolled in the Phase I safety and tolerability study, IMM-101-001. IMM-101-001 was a first-in-human (FIH), open-label, dose-escalation, intra-patient, placebo-controlled study, in adult patients with confirmed diagnosis of stage III or IV melanoma to evaluate the safety and tolerability of three doses of IMM-101 (further details are available in the FIH study clinical study report [CSR]).

In this long-term follow-up (LTF) study, IMM-101-008, IMM-101 (10 mg/mL) is administered as a single 0.1 mL intradermal injection every 4 weeks or as close to this interval as permitted due to practical or logistical considerations until death or withdrawal, unless such therapy is contraindicated, the patient does not wish to continue, or the study is terminated by the Sponsor.

The duration of this study is determined by the time to death or withdrawal of the last patient remaining in this study, hence the total duration of the study is not pre-determined.

This Statistical Analysis Plan (SAP) describes the intended statistical evaluation of the study data at the time of final study reporting based on the final study database.

This SAP is based on the study protocol (version 9.0, dated 18 October 2017, incorporating amendment numbers 1.0 to 8.0) and the final study case report form (CRF), version 4, dated 02 December 2012, the amended adverse event (AE) CRF version 3, dated 15 October 2013, and Post-Study Long Term Survival Status CRF version 1.0, dated 28 September 2015.

This SAP incorporates the original objectives outlined in the study protocol, the approved SAP dated 08 October 2015 and further amendments combining relevant data from the FIH study IMM-101-001 with the final study data for the LTF study IMM-101-008, in IMM-101-008-enrolled patients, thus providing an evaluation of the long-term safety profile of IMM-101 from first dosing in the FIH study through to last dosing in the LTF study, including the period between studies when patients were treated with IMM-101 under the Immodulon Named Patient Programme (NPP), when relevant data has been recorded in the LTF study CRF.

The FIH study results are reported in the CSR (date 01 March 2011), based on the final FIH study CRF version date 25 January 2010 and the final study database.

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

## 2. STUDY OBJECTIVE(S) AND ENDPOINT(S)

## 2.1 Study Objective(s)

The study objectives are,

- To determine the long-term safety profile of IMM-101 administered intradermally for extended use.
- To document the long-term clinical course of the patients previously enrolled in Study IMM-101-001.
- To monitor selected markers of tumour burden and immunological status.

The objective of this Statistical Analysis Plan (SAP) is to summarise the following outputs:

- Patient disposition
- Demographic characteristics
- Medical history
- Previous medications
- IMM-101 dose administration, time on study and exposure
- Injection site reactions
- Adverse events
- Overall Survival (OS)

The FIH and LTF combined data presentation objectives are to summarise the following outputs:

- Relevant medical events during the NPP (i.e. prior to entry to IMM-101-008)
- Anti-melanoma Cancer Therapies other than IMM-101 whilst on IMM-101 treatment
- IMM-101 administrations (from first dose of IMM-101 in the FIH study and including administrations during the LTF study)
- IMM-101 exposure
- Incidence and frequency of IMM-101-related treatment emergent AEs occurring following first dose
  of IMM-101 in the FIH study

## 2.2 Study Endpoint(s)

The Safety and Tolerability endpoints are:

- Local injection site tolerability
- Adverse Events with documentation of number, type and degree of toxicities as measured by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) v4.0 [1] where appropriate.

The Efficacy endpoints are:

- Overall survival
- Reduction in metastatic disease.

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Exploratory endpoints of change in markers of immune status are to be reported separately from the main endpoints of the study, and the analyses are not therefore described in this SAP.

#### 3. STUDY DESIGN

The LTF study is an open label long-term follow-up study of patients with melanoma who were previously enrolled in the Phase I FIH study IMM-101-001. The study consists of two phases; screening and enrolment, then treatment.

The screening period lasted up to 28 days to establish eligibility. Once confirmed as eligible, patients receive treatment every 4 weeks or as close to this interval as is permitted due to practical or logistical considerations until death or withdrawal, unless such therapy is contraindicated, the patient does not wish to continue or the study is terminated by the Sponsor. The dose interval can be modified at the discretion of the Investigator provided the minimum period between doses is no less than 14 days.

IMM-101 can be stopped if deemed necessary by the Investigator and/or patient, for example, due to intolerable injection site reactions. In the event of an injection site reaction of Grade 3 and above, at the discretion of the Investigator, patients may be administered a half dose of the study drug (i.e., a single 0.05 mL intradermal injection of IMM-101) or the time interval between doses may be increased. Patients can choose to withdraw from the study at any time and for any reason.

Protocol amendment 6.0 (dated 07 November 2014) allowed for a clinic telephone call to the patient to enquire about injection site reactions, adverse events, concomitant medications and any other concerns, if the patient does not attend for a study visit within a calendar month. Appropriate information is recorded in the CRF.

#### 4. PLANNED ANALYSES

At the time of final analysis for the study, descriptive summaries of the results of the study will be provided along with data listings of the final study database. Summary statistics or frequency tables will be provided, where appropriate.

Section 9 provides details of the descriptive statistics and TFL shells are included in Section 13.

No formal statistical analyses of the results are anticipated and hence no statistical inferences will be made.

Planned analyses as detailed in the protocol are as follows:

The evaluation of safety and tolerability will be summarised using the Safety population and will be based on local and systemic toxicities (including injection site tolerability) which will be presented over the treatment period in standard frequency tables, overall and by number, degree and type. Adverse Events will

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

be presented descriptively to include related adverse events, serious adverse events (SAEs), and adverse events leading to withdrawal or death. The frequency and severity of injection site reactions, and all other safety parameters will be summarised.

All patients will have received IMM-101 in the context of both the Phase 1 study and, for the majority, on a Named Patient basis; therefore all AEs in this long term follow up study will be regarded as treatment emergent.

Efficacy will be presented using the Safety population and will be assessed through documenting the long-term clinical course of the patients previously enrolled in Study IMM-101-001 in terms of OS. Reduction in metastatic disease will be listed only.

Variables for the exploratory endpoints will be analysed and reported separately to the main efficacy and safety endpoints of the study.

The protocol specified that OS will be presented from enrolment into this study, in addition to time from initial diagnosis and enrolment into study IMM-101-001. Time zero for the OS analysis in this study (IMM-101-008) will be based on the date of Day 0 in this study and analysis of OS taking into account time from initial diagnosis and first dosing day in Study IMM-101-001 will not be included in this SAP as not all patients completing the FIH study entered the LTF study.

In addition to the above planned presentations, non-serious adverse events in LTF study patients will be tabulated and treatment-related treatment emergent AEs will also be presented combining data in these patients, from both the FIH and LTF studies.

## 5. SAMPLE SIZE CONSIDERATIONS

Surviving patients from Study IMM-101-001 (EudraCT number: 2009-012447-42) who were continuing to receive IMM-101 on a Named Patient Programme (NPP) basis were invited to enrol into study IMM-101-008.

#### 6. ANALYSIS POPULATIONS

The Safety Population will comprise all patients who receive at least one dose of the study drug in the LTF study. All members of the Safety Population had previously been enrolled into the FIH study. Analysis of safety and tolerability endpoints and efficacy endpoints will be summarised on the Safety Population.

#### 7. GENERAL CONSIDERATIONS FOR DATA ANALYSES

In general, continuous data will be summarised using mean, standard deviation, minimum, median and maximum. The minimum and maximum will be recorded to the same number of significant figures as the

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

original data, whilst mean and median will be presented to 1 significant figure more than the original data, and standard deviation 2 significant figures more than the original data.

In summaries of categorical data, frequency counts and percentages will be used. Generally, percent will be displayed to one decimal place.

The time to event variable OS will be analysed using standard Kaplan-Meier techniques. The Kaplan Meier curve will be plotted and median (50%), 25% and 75% survival estimates reported with the corresponding 95% confidence intervals (CIs).

All analyses will be performed using SAS v 9.4 (or higher).

All tables, figures and listings (TFLs) will include titles, headers or footnotes which identify:-

- The analysis set on which the presentation is based.
- A description or title for the presentation (where combined data is presented from the FIH study and the LTF study, this will be indicated).
- The date and time the output was produced.
- A reference to the name and location of the file used to produce the output and the source of the data used (which may be a SAS dataset or another TFL).
- Reference to the analysis stage of the study data e.g. Final Analysis.

Listings which present data using repeating rows for a patient and/or visit will be presented in chronological date order (where applicable) with the repeating header information presented on the first new record for each repeating combination only, to facilitate readability.

All assessment data will be reported with the visit at which it was recorded, whether or not the visit falls inside the relevant window or not.

Tables and figures will be coded from Analysis Data Model (ADaM) format datasets. Listings will be coded from Study Data Tabulation Model (SDTM) datasets.

#### 8. DATA HANDLING CONVENTIONS

#### 8.1 Premature Withdrawal and Missing Data

Patients who withdraw early will be included in the analysis of safety and efficacy. Missing, unused and spurious data will be treated as such. No imputation methods will be applied, except for concomitant medication stop date as follows:

If the stop date for a medication is partially missing, it will be assumed to be a concomitant medication if, based on the partial information available, concomitant is not ruled out. Hence the date will be imputed to the end of the month/year, i.e. if day is unknown it will be set to the last day of the specified month, if day S:\Services\Immodulon\IMM-101-008\SMF\SAP\IMM-101-008\_SAPvFinal 1.1


**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

and month are unknown it will be imputed as 31<sup>st</sup> December. This imputation will be also used in the determination of whether the previous medication was stopped within 14 days prior to Day 0.

Date imputations will not be shown in data listings however, the flag based on imputed dates will be shown in the listings. Date imputations will be incorporated into tabulations of previous/concomitant medications.

## 8.2 Prior and Concomitant Therapy and Medical History Melanoma Therapies Coding

Each concomitant therapy recorded during the FIH and LTF studies will be categorised according to antimelanoma cancer therapy type as follows:

Chemotherapy

Cancer surgery (note: melanoma cancer surgeries only are included in this category)

Radiotherapy

Immunotherapy (other than IMM-101)

Radiofrequency ablation

Immunotherapy IMM-101.

Other categories may be considered, if relevant and mutually exclusive to the above.

A look-up table will be created containing the relevant verbatim term, dataset location and therapy code. Exploristics will supply dataset(s) in Excel format where verbatim terms for therapies contained in the previous and concomitant medications, and medical history datasets are listed, for allocation to one of the anti-melanoma cancer therapies codes by Immodulon. These will be medically reviewed by Immodulon and approved prior to issue of final TFLs. Listings will include the assigned categories, where allocated.

All concomitant therapy groupings with the exception of immunotherapy IMM-101 will be included in the tabulation of anti-cancer (melanoma-related) therapies. Therapies included will be all therapies given after first dose of IMM-101 in the FIH study, including co-medication during NPP treatment (recorded as medical history since leaving the FIH study) and during the LTF study.

## 8.3 Derived and Transformed Data

As age was not collected it will be derived using the patient's date of birth and date of consent. The derivation will be

Age (years) = integer part of ((patient informed consent date - date of birth + 1)/365.25).

Note that the full date of birth will be used in the calculation, but only year of birth will be listed. Patient initials will not be listed.

## **Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Time since initial diagnosis of current presentation, time since excision of primary lesion, time since excision of sentinel node and time since regional lymph node resection will be derived in years as follows;

Time since initial diagnosis of current presentation (years) = (Day 0 - date of initial diagnosis of current presentation + 1)/ 365.25

Time since excision of primary lesion (years) = (Day 0 - date of excision of primary lesion + 1)/365.25.

Time since excision of sentinel node (years) = (Day 0 - date of excision of sentinel node + 1)/365.25 and missing if not excised.

Time since regional lymph node resection (years) = (Day 0 - date of regional lymph node resection + 1)/365.25 and missing if not resected.

The relevant time variable above will be reported to 1 decimal place, but calculated using all accuracy available in the data. If any dates are partial, i.e. day number missing, the time variable will be calculated using month and year only and if day and month missing, the time variable will be calculated using year only as follows:

- If only month and year are present (MMYYYY): Time since Event = (Day 0 Event date +1) / 365.25;
- If only year is present (YYYY): Time since Event = (Day 0 Event date) +1 / 365.25.

The total number of pre-study doses of IMM-101 received (since the completion of study IMM-101-001) will be calculated for each patient.

Exposure during the IMM-101-008 study will be summarised by time on study in years and overall exposure in months, which will be derived using:

**Time on study (years)** = (date of study completion (i.e. death on study)/date of withdrawal) - Day 0 + 1/365.25.

Overall study drug exposure (months) = (date of last dose - date of first dose in study IMM-101-008 + 1)/30.4375.

Overall exposure of IMM-101 (FIH and LTF study combined) will be derived using: (date of last dose in study IMM-101-008 – date of first dose in study IMM-101-001 + 1)/30.4375.

On-study dosing will be summarised using the total number of doses on study:

**Total no. doses on study** = (Total number of IMM-101 doses whilst on the LTF study by totalling the doses (full or part doses counted as 1 dose) recorded in the CRF.

Time elapsed since previous dose (for on-study administration of IMM-101) will be derived using;

S:\Services\Immodulon\IMM-101-008\SMF\SAP\IMM-101-008 SAPvFinal 1.1


**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

**Time elapsed since previous dose (days)** = (date of current dose - date of previous dose + 1).

A **dose change flag** (Dose changed from previous dose, I = increased, D = decreased) will be used to record any escalation or reduction in dose received between consecutive visits. If the dose has remained consistent compared to previous dose, this flag will remain unoccupied.

Time to event analysis will be performed on OS which will be calculated in years, from Day 0 in study IMM-101-008 using;

Overall Survival (years) = (date of death - Day 0 + 1)/365.25OR (censored date - Day 0 + 1)/365.25

See Section 10 for additional information.

Adverse events and medical history will be coded using MedDRA v 18.0 (or higher). MedDRA will be used to create System Organ Class (SOC) and Preferred Term (PT) variables.

A flag (Stopped >14 days prior) will be created for previous medications which were taken and stopped before 14 days prior to the end of screening procedures (i.e. Day 0) based on the medication end date and date of Day 0.

Previous and concomitant medications and significant medical history since completing the FIH study will undergo coding for anti-melanoma cancer treatments, see Section 8.2.

Note: Derived variables recorded in the unit of months or years will be reported to 1 decimal place, derived variables recorded in the unit of days will be reported to whole numbers only. Age will be reported to whole years only.

Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

#### 9. DESCRIPTIVE STATISTICS

## 9.1 Disposition of Patients

The number and percentage of patients meeting all inclusion criteria, completing (i.e. dying) and withdrawing will be summarised (Table 1), along with reasons for death and withdrawal from study.

## 9.2 Demographic and Baseline Characteristics

Patient demographics will be presented in Table 2.

Specific melanoma medical history is summarised in Table 3a which includes a summary of any lesions present during the screening period, by location. The number and percentage of patients with significant medical history (non-melanoma specific) since completion of study IMM-101-001 categorised by SOC and PT using MedDRA v 18.0 (or higher) will be presented in Table 3b.

Data summaries of pre-study administration by IMM-101 dose received since completing study IMM-101-001 can be found in Table 4. Pre-existing injection site reactions, and any history of severe local reactions following previous administration(s) of IMM-101 will be summarised as a frequency table (Table 5).

Previous medications are prescription/non-prescription drugs, vitamins, drugs of abuse and dietary supplements taken and stopped within 14 days prior to Day 0. Any previous medications stopped before 14 days prior to Day 0 will be identified with a flag in the listings. Any medications, including vitamins, and dietary supplements ongoing or started on/after Day 0 and surgical procedures are defined as Concomitant Therapies.

The incidence of patients receiving at least one anti-melanoma cancer therapy other than IMM-101 and ongoing or started on or after the first dose of IMM-101 in the FIH study will be summarised for the FIH and LTF studies combined. Overall incidence will be summarised as well as by therapy type and therapy verbatim term (i.e. description of treatment given). IMM-101 treatments and non-melanoma cancer therapies will not be included in the tabulation (Table 6). Concomitant treatments received during the FIH study were recorded in the FIH study CRF. Treatments for relevant medical history including relevant radiotherapy, cancer surgery, chemotherapy and immunotherapy received following completion of the FIH study and prior to entry to the LTF study and any medications taken within 14 days prior to the LTF study screening visit as well as concomitant treatments received after entry to the LTF study are recorded in the LTF study CRF.

#### 9.3 Study Treatment, Exposure and Safety Outputs

An on-study administration table (Table 7) will show the number and percentage of patients who receive study drug and whether full dose or reduced dose was administered, summarised by visit. In these

# Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

presentations, the denominator for the calculation of percentages at each visit will be based on the number of patients available at each visit who provide a response.

A line graph for each patient will be plotted to visually display any variation in doses of IMM-101 (in mg) by time, during the LTF study. This will be presented in the form of a panel plot (Figure 1a) on standard axes for each patient. Each dose will be marked by an 'X' on the plot. In addition, a panel plot (Figure 1b) will be presented including all IMM-101 doses received from the first dose in the FIH study, to the last dose in the LTF study, inclusive including those taken whilst the patient was being treated in the NPP, in a similar manner.

Exposure, to include the time on LTF study in years, overall LTF study drug exposure (months) and total no. doses on study, will be summarised in Table 9a.

Overall exposure to IMM-101 from first dose in the FIH study to last dose in the LTF study inclusive will be summarised in Table 9b.

Summaries of adverse events will include the number of adverse events and the proportion of patients experiencing at least one adverse event. If an individual patient has more than one AE at a given level of classification the patient will be counted only once at the given level of classification but each event will be counted within the number of events associated with that level of classification.

All patients will have received IMM-101 in the context of both the Phase 1 study IMM-101-001, and, for the majority, during the NPP; therefore all AEs in this long-term follow-up study will be regarded as treatment-emergent.

Table 10a includes the incidence and frequency of all TEAEs, treatment emergent treatment-related AEs, treatment emergent SAEs, Serious treatment-related TEAEs, TEAEs resulting in withdrawal or death and AEs of NCI CTCAE Grade ≥ 3.

Frequency summaries of treatment emergent adverse events by SOC and PT using MedDRA v 18.0 (or higher) will be included overall (Table 10b) and repeated to capture:-

- Treatment emergent adverse events of NCI Grade ≥3 (Table 10c)
- Treatment emergent, IMM-101-related, adverse events: AEs that are definitely, probably or possibly related to study drug or with an unknown relationship (Table 10d)
- Treatment emergent, SAEs (Table 10e)
- Treatment emergent adverse events leading to withdrawal or death (Table 10f).
- Treatment emergent non-serious adverse events (Table 10g).

Additionally, long term safety will be evaluated by combining treatment related adverse event experience in the FIH study through to the end of the LTF study by summarising treatment emergent treatment-related adverse events (IMM-101-001 and IMM-101-008 Combined) (Table 10h).

**Exploristics Limited** Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Where it is not applicable to grade an AE using NCI CTCAE grade, it will be excluded from the summary of NCI Grade 3 and above AEs. Any AEs with missing grades, however, will be included, based on a worst-case approach.

On-study injection site reactions are summarised over the treatment period by visit in Table 11.

Urine Pregnancy Test Results and blood samples for immunological markers will be listed but not summarised.

All safety data will be listed.

Any comments recorded as free text in the CRF will be listed.

#### 10. ANALYSIS CORRESPONDING TO THE STUDY OBJECTIVES

Overall Survival (OS) is defined as the time from a patient's date of Day 0 until date of death. Patients still alive will be censored at withdrawal from the study or at last known date alive if later (where patients have consented to follow-up for overall survival outcome, after they have withdrawn from the study). If consent has been provided by the patient, the patient's final outcome will be included if death and if alive, the patient will have censored outcome at the date last known to be alive.

Post-study survival status after withdrawal from the study, for any withdrawn patients, will be recorded on a separate Post-study Long Term Survival Status CRF, and these data will be included in the analysis and data listings, as described above.

The patient's death is recorded as the date of study completion on CRF page 18 and if after withdrawal from the study, the date of death recorded on the Post-study CRF.

A patient without a death date will be censored in the analysis at the last date known to be alive providing their consent was obtained. Patients withdrawing from the study without consent for further follow up will be censored for survival at the date of their withdrawal from the study (recorded on CRF page 18).

Overall Survival will be summarised by Kaplan-Meier curves. Median, 25% and 75% survival estimates as well as associated 95% CIs will be reported in Table 8 and Figure 2.

SAS procedure output for the OS analysis will be included as an appendix to the CSR.

**Exploristics Limited**Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

The changes in metastatic disease compared with previous assessment (as measured via CT or MRI scan) recorded at the discretion of the investigator, will be presented over the treatment period in data listings only (Listing 11).

#### 11. PROTOCOL DEVIATIONS AND DEVIATIONS FROM PLANNED ANALYSIS

Protocol deviations will be reported separately, based on the study protocol deviations log maintained by Immodulon, and included in the CSR directly.

Any substantive deviations from the planned data presentations and analysis described in this SAP will be documented along with reason for change, in the CSR.

Overall survival will be calculated from the date of Day 0, not enrolment into the study, as the enrolment period may be up to 28 days long.

#### 12. REFERENCES

[1] Cancer Therapy Evaluation Program, Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0, DCTD, NHI, DHHS, 28 May 2009.

Exploristics Limited Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

## 13. ATTACHMENTS

# 13.1 Table of Contents for Data Display Specifications

| Tables | |
|---|---|
| 1 | Summary of Patient Disposition |
| 2 | Demographics |
| 3a | Melanoma Specific Medical History |
| 3b | Significant Medical History since Completion of Study IMM-101-001 |
| 4 | Pre-study IMM-101 Administration Since Completion of Study IMM-101-001 |
| 5 | Pre-Existing Injection Site Reaction(s) |
| 6 | Summary of Anti-melanoma Cancer Therapies other than IMM-101 Whilst on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined) |
| 7 | On-Study IMM-101 Administration |
| 8 | Overall Survival |
| 9a | Exposure |
| 9b | Time on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined) |
| <b>10</b> a | Summary of Treatment Emergent Adverse Events |
| 10b | Treatment Emergent Adverse Events |
| <b>10</b> c | Treatment Emergent Adverse Events with NCI CTCAE Grade ≥ 3 |
| <b>10</b> d | Treatment Emergent Adverse Events Related to IMM-101 |
| <b>10</b> e | Treatment Emergent Serious Adverse Events |
| 10f | Treatment Emergent Adverse Events Leading to Withdrawal or Death |
| 10g | Treatment emergent Non-serious Adverse Events |
| 10h | Treatment-related Treatment Emergent Adverse Events (IMM-101-001 and IMM-101-008 Combined) |
| 11 | On-Study Injection Site Reaction(s) |

| | • | | | |
|---|-----|-----|---|----|
| | | • | n | gs |
| L | .13 | SLI | | 23 |

| 1 | Patient Disposition |
|------|-----------------------------------------------------------------------|
| 2 | Demographics |
| 3a | Inclusion/Exclusion Questions |
| 3b | Inclusion/Exclusion Criteria |
| 3c | Inclusion/Exclusion Criteria Confirmation |
| 4ai | Melanoma Specific Medical History |
| 4aii | Melanoma Specific Medical History Continued |
| 4b | Significant Medical History since Completion of Study IMM-101-001 |
| 5 | Pre-Existing Injection Site Reaction(s) Assessed at Screening |
| 6 | Screening Urine Pregnancy Test Results |
| 7 | Disease and Treatment History at Screening |
| 8a | Previous Medications |
| 8b | Concomitant Therapies |
| 9 | Previous IMM-101 Administration Since Completion of Study IMM-101-001 |
| 10 | On-Study IMM-101 Administration |
| 11 | On-Study Disease Assessment |

**Exploristics Limited** 

2

#### Clinical Study Identifier: IMM-101-008 **Adverse Events** 12 On-Study Injection Site Reaction(s) 13 Concomitant Medication and Adverse Event Checks 14 Study Visits and Visit Checklists 15 Blood Sample for Immunological Markers 16 Post-Study Long Term Survival Status **17** Additional Comments Recorded 18 **Figures** Panel Plot of On-Study IMM-101 Doses by Patient **1**a All IMM-101 Dosing Administrations (IMM-101-001 and IMM-101-008 Combined) 1b

Kaplan Meier Curve of Overall Survival

Identifier: EXP12002

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

(응)

N = xx

## 13.2 Data Display Specification

Final Analysis

Protocol: IMM-101-008

Analysis Population: All patients

Page x of y

# Table 1 Summary of Patient Disposition

| | 1/1 — XX | ( 0 ) |
|---|---|---|
| Number of patients who entered the study | XX | |
| Number of patients in the safety population | XX | (xx.x) |
| Number of patients who met all Inclusion/Exclusion criteria | XX | (xx.x) |
| Number of patients who died on study | XX | (xx.x) |
| Reason for death | | |
| Adverse event/unacceptable toxicity | XX | (xx.x) |
| Other: Death due to disease progression | XX | (xx.x) |
| Number of patients who withdrew from the study | XX | (xx.x) |
| Reason for Withdrawal | | |
| Adverse event/unacceptable toxicity | XX | (xx.x) |
| Patient request/withdrawal of consent | XX | (xx.x) |
| Investigator decision | XX | (xx.x) |
| Did not meet inclusion/exclusion criteria | XX | (xx.x) |
| Pregnancy | XX | (xx.x) |
| Non-compliant | XX | (xx.x) |
| Other | XX | (xx.x) |

Note: Percent is based on the total number of patients in the Safety Population.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table1.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Completion date is date of death. Death reasons are recorded in categories stated.

Note to programmer: The number of patients who met all Inclusion/Exclusion criteria is based on response from page 12 of the CRF

Table 2

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

| Demographics | |
|-------------------------------------|------------|
| | N = xx (%) |
| Age at informed consent (yrs) | |
| N | XX |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | xx |
| Gender (%) | N |
| Female | xx (xx.x) |
| Male | xx (xx.x) |
| If Female: Child-bearing status (%) | N |
| Post-menopausal | xx (xx.x) |
| Surgically sterile | xx (xx.x) |
| Childbearing potential | xx (xx.x) |
| Unknown | xx (xx.x) |
| Race/ethnicity (%) | N |
| Black/Afro-Caribbean | xx (xx.x) |

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

| White/Caucasian Asian Other | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
|-----------------------------|-------------------------------------|
| Height (cm) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. | XX |
| Max. | xx |
| WHO performance status (%) | N |
| 0 | xx (xx.x) |
| 1 | xx (xx.x) |
| 2 | xx (xx.x) |
| 3 | xx (xx.x) |
| 4 | xx (xx.x) |

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Note: Percent is based on the number of patients who provided a response for each criteria.

Note: Age at informed consent derived using: Age (years) = integer part of ((patient informed consent date - date of birth + 1)/365.25). Full date of birth is used in the calculation, but only year of birth is listed.

Note: WHO performance status assessment

0=Asymptomatic, 1=Symptomatic but completely ambulatory, 2=Symptomatic <50% in bed during the day, 3=Symptomatic >50% in bed but not bedbound, 4=Bedbound.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table2.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 3a Melanoma Specific Medical History

| | N = XX (%) |
|--------------------------------------------------------------|------------|
| Time since initial diagnosis of current presentation (years) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | xx.x |
| Min. | xx |
| Max. | XX |
| Time since excision of primary lesion (years) | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | XX |
| Time since excision of sentinel node (years) | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | XX |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

| Max. | xx |
|---------------------------------------------------------------|----------|
| Time since resection of regional lymph node resection (years) | |
| N | xx |
| Mean | xx.x |
| SD | XX.XX |
| Median | XX.X |
| Min. | xx |
| Max. | xx |
| Stage of disease (%) | N |
| Stage III a | xx(xx.x) |
| Stage III b | xx(xx.x) |
| Stage III c | xx(xx.x) |
| Stage IV | xx(xx.x) |
| Unknown | xx(xx.x) |
| Other | xx(xx.x) |
| Primary lesion thickness (T type) (mm) | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |
| Median | XX.X |
| Min. | XX |
| Max. | XX |
| Presence of lymph node metastases (N type) (%) | N |
| Yes | xx(xx.x) |
| No | xx(xx.x) |
| Unknown | xx(xx.x) |

# **Exploristics Limited**

Identifier: EXP12002 Clinical Study Identifier: IMM-101-008

| Current lesions (%) | N |
|-----------------------------------|----------|
| Yes | xx(xx.x) |
| No | xx(xx.x) |
| Unknown | |
| If Yes: Location of lesion(s) (%) | N |
| Location 1 | xx(xx.x) |
| Location 2 | xx(xx.x) |
| Location n | xx(xx.x) |

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Note: As patients may have more than one lesion in various locations they can be included in more than one location category.

Note: Percent is based on the number of patients who provided a response for each criteria.

Note: Time (years) since variables are calculated from Day 0 + 1 and divided by 365.25.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table3a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Locations listed under PELOC e.g. Lung.

Note to programmer: If stage is other and more information is provided include it in the other description or as a footnote.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

Note to programmer: Please add footnote if any 'time since' variables contain partial missing dates, see SAP section 8.2: Where day and month are not known for either date, calculation is based on year alone: Time since event (years) = (Year of Day 0 - Year of event) + 1/365.25, likewise if day is not known for either date, calculation is based on month and year only

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Table 3b

Significant Medical History since Completion of Study IMM-101-001

System Organ Class

| Preferred Term | N = xx (%) |
|---|---|
| Significant or clinically relevant medical history since completion of study IMM-101-001? | N |
| Yes | xx(xx.x) |
| No | xx(xx.x) |
| Unknown | xx(xx.x) |
| If Yes: | |
| System Organ Class | N |
| Preferred Term 1 | xx(xx.x) |
| Preferred Term 2 | xx(xx.x) |
| Preferred Term n | xx(xx.x) |

Note: Medical History is coded using MedDRA version xx.x.

Note: Percent is based on the number of patients in the Safety Population.

 $\label{lem:code:s:Services} Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table3b.sas \ ddmmmyy:hh:mm:ss \ ddmmmyy:hh:mm:sd \ ddmmmyy:hh:mm:sd$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Please add relevant MedDRA version number in note to reflect version used at time of coding.

Note to programmer: Sort SOC and PT by decreasing incidence.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Table 4
Pre-study IMM-101 Administration Since Completion of Study IMM-101-001

| | N = xx (%) |
|---|---|
| Any IMM-101 administration(s) since the completion of the Phase 1 study IMM-101-001(%) Yes No | xx(xx.x)<br>xx(xx.x) |
| Number of patients who received at least 1 dose of: (%) | |
| xx.x mg | xx(xx.x) |
| xx.x mg | xx(xx.x) |
| xx.x mg | xx(xx.x) |
| Total number of doses administered over all patients at dose of: | |
| xx.x mg | XX |
| xx.x mg | XX |
| xx.x mg | XX |
| Total number of doses administered pre-study | xx |
| Total number of doses received per patient | |
| N | XX |
| Mean | XX.X |
| SD | XX.XX |

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

| Median | XX.X |
|--------|------|
| Min. | XX |
| Max. | XX |

Note: Percent is based on the number of patients who provided a response for each criteria.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table4.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 5 Pre-Existing Injection Site Reaction(s)

| N=xx (%) |
|-----------|
| N |
| N |
| xx(xx.x) |
| xx(xx.x) |
| xx (xx.x) |
| N |
| xx(xx.x) |
| xx(xx.x) |
| xx(xx.x) |
| xx(xx.x) |
| xx (xx.x) |
| N |
| xx(xx.x) |
| xx(xx.x) |
| xx(xx.x) |

Note: Percent is based on the number of patients who provided a response for each criteria.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table5.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

#### Table 6

Summary of Anti-melanoma Cancer Therapies other than IMM-101 Whilst on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined) N=XX

| Number of patients with at least one other anti-cancer | v | (xx.x) |
|--------------------------------------------------------|---|--------|
| therapy | X | (XX.X) |
| Cancer Surgery | Х | (xx.x) |
| XXXX | X | (xx.x) |
| XXXX | X | (xx.x) |
| Chemotherapy | X | (xx.x) |
| XXXX | X | (xx.x) |
| Immunotherapy | X | (xx.x) |
| XXXX | X | (xx.x) |
| Radiotherapy | X | (xx.x) |
| XXXX | Х | (xx.x) |
| Radiofrequency Ablation | X | (xx.x) |

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

X = XX

Note: Anti-melanoma cancer Therapies include melanoma-related surgery, chemotherapy, radiotherapy, radiofrequency ablation and non-IMM-101 immunotherapy treatments ongoing or started on/after the first dose of IMM-101 in study IMM-101-001, including therapies during NPP (recorded as medical history since leaving study IMM-101-001) and during IMM-101-008.

Note: Therapies are counted once per therapy type per patient hence duplicates are not included in the table.

Note: Percent is based on the total number of patients in the Analysis Population.

XXXX

Note: MedDRA preferred terms are reported for procedures reported with AEs. Otherwise, verbatim terms are reported. Preferred Term is coded using MedDRA version 18.1

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table6.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxx.sas7bdat, S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxxx.sas7bdat,

S:\Services\Immodulon\IMM-101-008\DataManagement\DataEntry\Coding Files\cancer coding lookup xx xxx xxxx.sas7bdat,

Note to programmer: Please update data footnote with appropriate file directory. Please sort by decreasing incidence at therapy type and treatment level. Non-cancer treatments and immunotherapy IMM-101 will be excluded from this table.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Table 7
On-Study IMM-101 Administration

| | Visit 1 | Visit N |
|----------------------------|----------|----------|
| | N | N |
| IMM-101 dose administered? | | |
| No | xx(xx.x) | xx(xx.x) |
| Yes | xx(xx.x) | xx(xx.x) |
| If Yes: | | |
| Full dose (1 mg) | xx(xx.x) | xx(xx.x) |
| Reduced dose (<1 mg) | xx(xx.x) | xx(xx.x) |

Note: The percent will be based on the number of patients available at each visit who provide a response.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table7.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Where 'Visit N' appears add additional columns as required. If too many Visits for columns create sets of rows for each visit number.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

# Table 8 Overall Survival

| Total number of patients | XX |
|-------------------------------|----------------------------|
| Number of deaths | XX |
| Number of censored events | xx |
| Median survival time (95% CI) | xx.x ( $xx.xx$ , $xx.xx$ ) |
| 25% survival time (95% CI) | xx.x (xx.xx, xx.xx) |
| 75% survival time (95% CI) | xx.x (xx.xx, xx.xx) |

Note: The summary statistics for survival time have been derived based on the Kaplan-Meier product limit survival estimates.

Note: Overall survival (years) is calculated as ((date of death or censored date) - Day 0 + 1)/365.25.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table8.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Table 9a

Analysis Population: Safety Population

| Exposure | |
|-------------------------------------------|--------|
| 2 111 1 | N = xx |
| Time on study (years) | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | xx |
| Overall study drug exposure (months) | |
| N | xx |
| Mean | XX.X |
| SD | xx.xx |
| Median | xx.x |
| Min. | xx |
| Max. | xx |
| Total no. IMM-101 doses received on study | |
| N | xx |
| Mean | xx.x |
| SD | xx.xx |
## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Median xx.x Min. xx Max. xx

Note: Time on study (years) = (date of completion (i.e. death on study)/date of withdrawal - Day 0 + 1)/365.25.

Overall Exposure (months) = (date of last dose - date of first dose in study IMM-101-008 + 1)/30.4375.

Total number of doses received = sum of the doses (full or part doses counted as 1 dose) received, as reported in the CRF.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table9a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Decimal places for continuous data summaries are based on the variable recorded in the data being to zero decimal places. If the decimal places recorded are increased in the data then increase decimal places for mean, median, SD, min and max in the table accordingly.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

Table 9b

Time on IMM-101 Treatment (IMM-101-001 and IMM-101-008 Combined)

Overall study drug exposure (months)

 N
 X

 Mean
 xx.xx

 StD
 xx.xxx

 Median
 xx.xx

 Min.
 xx.x

 Max.
 xx.x

Note: Overall study drug exposure is derived as follows:

Overall study drug exposure (months) = (date of last dose in study IMM-101-008 - date of first dose in study IMM-101-001 + 1)/30.4375.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\ Table9b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxx.sas7bdat,

S:\Services\Immodulon\IMM-101-001\RawData SDTM\xxxxxx.sas7bdat,

S:\Services\Immodulon\IMM-101-008\SDTM\ xxxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Table 10a
Summary of Treatment Emergent Adverse Events

| | N = xx (%) |
|---|---|
| Number of patients with treatment emergent adverse events (%) | xx(xx.x) |
| Number of treatment emergent adverse events | XX |
| Number of patients with treatment emergent adverse events related to the study drug (%) | xx(xx.x) |
| Number of treatment emergent adverse events related to the study drug | XX |
| Number of patients with serious treatment emergent adverse events (%) | xx(xx.x) |
| Number of serious treatment emergent adverse events | XX |
| Number of patients with serious treatment emergent adverse events relating to the study drug (%) | xx(xx.x) |
| Number of serious treatment emergent adverse events relating to the study drug | XX |
| Number of patients with treatment emergent adverse events leading to withdrawal or death (%) | xx(xx.x) |
| Number of treatment emergent adverse events leading to withdrawal or death | XX |
| Number of patients with treatment emergent adverse events of NCI CTCAE $\geq$ Grade 3 (%) | xx(xx.x) |
| Number of treatment emergent adverse events of NCI CTCAE ≥ Grade 3 | XX |

Note: Treatment emergent AEs are all those reported during the study. Related AEs are defined as events that are definitely, probably or possibly related to study drug or with an unknown relationship.

Note: CTCAE - Common Toxicity Criteria for Adverse Events CTCAE decode.

Note: Percent is based on total number of patients in the Safety Population.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10b Treatment Emergent Adverse Events

| System Organ Class/ | |
|---------------------------------------------------------------|-----------|
| Preferred Term | N = XX |
| | n(%) m |
| Number of patients with treatment emergent adverse events (%) | xx(xx.x) |
| Total Number of treatment emergent adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

#### Table 10c

Treatment Emergent Adverse Events with NCI CTCAE Grade ≥ 3

| System Organ Class/ Preferred Term | N = xx<br>n(%) m |
|---|---|
| Number of patients with treatment emergent adverse events of NCI CTCAE $\geq$ Grade 3 Total Number of treatment emergent adverse events of NCI CTCAE $\geq$ Grade 3 | xx (xx.x)<br>xx |
| System Organ Class Preferred Term | n(xx.x) m<br>n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

Note: Common Toxicity Criteria for Adverse Events CTCAE decode. 1. Mild, 2. Moderate, 3, Severe, 4. Life Threatening, 5. Death

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10c.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10d Treatment Emergent Adverse Events Related to IMM-101

| System Organ Class/ | N = XX |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with treatment emergent, related adverse events (%) | xx(xx.x) |
| Total Number of treatment emergent, related adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study. Related AEs are defined as events that are definitely, probably or possibly related to study drug or with an unknown relationship.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10d.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10e Treatment Emergent Serious Adverse Events

| System Organ Class/ | N = xx |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with serious, treatment emergent adverse events (%) | xx(xx.x) |
| Total Number of serious, treatment emergent adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

 $\label{thm:ss} \textbf{Code: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash Analysis\backslash Development\backslash Code\backslash Table 10e.sas \ ddmmmyy: hh:mm:ss} \\$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

#### Table 10f

Treatment Emergent Adverse Events Leading to Withdrawal or Death

| System Organ Class/ | N = XX |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with treatment emergent adverse events leading to withdrawal or death (%) | xx(xx.x) |
| Total Number of treatment emergent adverse events leading to withdrawal or death | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; <math>m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted

under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported during the study.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10f.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Table 10g Treatment Emergent Non-serious Adverse Events

| System Organ Class/ | |
|---|---|
| Preferred Term | N = XX |
| | n(%) m |
| Number of patients with treatment emergent non-serious adverse events (%) | xx(xx.x) |
| Total Number of treatment emergent non-serious adverse events | XX |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with a non-serious AE; <math>m = number of non-serious AEs.

Hence if a patient has multiple non-serious AEs only one occurrence per person will contribute to 'n', but all occurrences will

be counted under  $\mbox{'m'}$  as this is the total number of non-serious events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent non-serious AEs are all those reported during the study.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table10g.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

Note to programmer: Please add relevant version number in MedDRA note to reflect version used at time of coding

Note to programmer: All non-serious AEs are to be excluded from this summary table.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

#### Table 10h

Treatment-related Treatment Emergent Adverse Events (IMM-101-001 and IMM-101-008 Combined)

| System Organ Class/ | N = xx |
|---|---|
| Preferred Term | n(%) m |
| Number of patients with treatment-related treatment emergent adverse events (%) | xx(xx.x) |
| Total Number of treatment-related treatment emergent adverse events | xx |
| System Organ Class | n(xx.x) m |
| Preferred Term | n(xx.x) m |

Note: n = number of patients with an AE; m = number of AEs.

Hence if a patient has multiple AEs only one occurrence per person will contribute to 'n', but all occurrences will be counted under 'm' as this is the total number of events recorded.

Note: Preferred Term and System Organ Class are coded using MedDRA version 18.1.

Note: Percent is based on the total number of patients in the Safety Population.

Note: Treatment emergent AEs are all those reported at/after first IMM-101 dosing in study IMM-101-001. Related AEs are defined as AEs that are definitely, probably or possibly related to study drug or with an unknown relationship.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\ Table10h.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Data: S:\Services\Immodulon\IMM-101-001\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory. Note to Programmer: Order by most common (by incidence) SOC and PT within SOC.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

Table 11
On-Study Injection Site Reaction(s)

| | Visit 1<br>N = xx (%) | Visit 2<br>N = xx (%) | Visit N<br>N = xx (%) |
|---|---|---|---|
| Is the injection site reaction from previous IMM-101 dose(s) visible? | N | N | N |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| If visible, are daily activities affected? | N | N | N |
| Not at all | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Slightly | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderately | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Quite badly | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intolerably | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Worsening with repeated doses of IMM-101? | N | N | N |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Sure | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Wound care required? | N | N | N |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Percent are based on the number of patients available at each visit who provided a response.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Table11.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Where 'Visit N' appears add additional columns as required, or reverse rows and columns if visits large in number, so rows become visits and variables are in the columns.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

# Listing 1 Patient Disposition

| Unique<br>Patient ID | Consent Date<br>(DD-MM-<br>YYYYTHH:MM) | Versio<br>n<br>Number | Off-Study<br>Date<br>(DD-MM-YYYY) | Off-<br>Study<br>Status | Time on<br>Study<br>(years) | Overall<br>Study<br>drug<br>exposure<br>(months) | Total no. IMM- 101 Doses receiv ed on Study | Reason<br>for<br>Completio<br>n (death)<br>or<br>Withdrawa | All adverse events<br>followed for at<br>least 30 days<br>after study<br>completion/withdra<br>wal | Principal Investiga tor Sign off Date (DD-MM- YYYY) |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | xxxxx | XX | XX | XX | xxxxx | xxxxx | DD-MM-<br>YYYY |
| XXXXX | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | XXXXX | XX | XX | XX | XXXXX | xxxxx | DD-MM-<br>YYYY |
| XXXXX | DD-MM-YYYY HH:MM | xx | DD-MM-YYYY | XXXXX | XX | XX | XX | XXXXX | xxxxx | DD-MM-<br>YYYY |
| XXXXX | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | XXXXX | XX | XX | XX | XXXXX | xxxxx | DD-MM-<br>YYYY |
| xxxxx | DD-MM-YYYY HH:MM | xx | DD-MM-YYYY | XXXXX | xx | xx | xx | xxxxx | xxxxx | DD-MM- |
| xxxxx | DD-MM-YYYY HH:MM | XX | DD-MM-YYYY | XXXXX | XX | XX | XX | xxxxx | xxxxx | YYYY<br>DD-MM-<br>YYYY |

Note: Time on study (years) = (date of completion (i.e. death on study)/date of withdrawal - Day 0 + 1)/365.25.

Overall Exposure (months) = (date of last dose - date of first dose in study IMM-101-008 + 1)/30.4375.

Total number of doses received = sum of the doses (full or part doses counted as 1 dose) received, as reported in the CRF.

Note: The trial was terminated in Dec-2018 as no further meaningful data was being collected nor was likely to be collected in the future.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing1.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Off-Study Status should be either 'Completed Study - patient died' or 'Withdrew'.

Note to Programmer: Where applicable, separate date from time using a space.

Note to Programmer: Status at completion/withdrawal: If reason is AE/unacceptable toxicity, Investigator decision or Patient did not meet INC/EXC criteria, please include specify text. If reason is other please include reason/description where applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 2
Demographics

| Unique<br>Patient<br>ID | Year of<br>Birth<br>(YYYY) | Age at Informed Consent (years) | Race/<br>Ethnicity | Gender | Child-<br>bearing<br>Status | Height<br>(cm) | WHO<br>Performance<br>Status |
|---|---|---|---|---|---|---|---|
| ' | | | | | | | |
| XXXXX | YYYY | XX | XXXXX | XXXXX | XXX | XXX | X |
| XXXXX | YYYY | XX | XXXXX | XXXXX | XXX | XXX | X |

Note: Age at informed consent will be derived using; Age (years) = integer part of ((patient informed consent date - date of birth + 1)/365.25).Note: Full date of birth is used in the calculation, but only year of birth is listed.

Note: WHO performance status assessment

0=Asymptomatic, 1=Symptomatic but completely ambulatory, 2=Symptomatic <50% in bed during the day, 3=Symptomatic >50% in bed but not bedbound, 4=Bedbound.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing2.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: If Race/ethnicity was recorded as 'Other' on the CRF then the response provided should be listed.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Not Applicable

# Listing 3a Inclusion/Exclusion Questions

| Question<br>Number | Inclusion/<br>Exclusion<br>Criteria | Question |
|---|---|---|
| 1 | Inclusion | Were previously enrolled in Study IMM-101-001. |
| 2 | Inclusion | Give consent to make their disease and treatment history for the intervening period between their completion of Study IMM-101-001 and enrolment in this study available to the Sponsor. |
| 3 | Inclusion | Give signed informed consent for participation in the study. |
| 1 | Exclusion | Female patient of child-bearing potential who is not, in the opinion of the Investigator, using an approved method of birth control (e.g., physical barrier [patient and partner], contraceptive pill or patch, spermicide and barrier, or intrauterine device [IUD]). Those patients that utilise hormonal contraceptives must have used the same method for at least three months before additional barrier contraception (as described above) is discontinued from being used concomitantly with the hormonal contraception. Patient of non-child-bearing potential are defined as having 12 month amenorrhoea or are surgically sterile. |
| 2 | Exclusion | Female patient who is pregnant, breast feeding or planning a pregnancy during the course of the study. A pre-treatment urine pregnancy test measuring human chorionic gonadotrophin (HCG) must be negative. |
| 3 | Exclusion | Patient is unable or unwilling to comply with the protocol. |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing3a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Listing 3b
Inclusion/Exclusion Criteria

| Unique<br>Patient ID | Date of<br>Collection<br>(DD-MM-YYYY) | Question<br>Number | Inclusion/<br>Exclusion<br>Criteria | Criteria<br>Met?<br>(Y/N) |
|---|---|---|---|---|
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| XXXXX | DD-MM-YYYY | XX | XXXXX | XX |
| xxxxx | DD-MM-YYYY | XX | xxxxx | XX |

Note: Reference Listing 3a for Inclusion/Exclusion Criteria Questions

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing3b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Inclusion / Exclusion criteria will be used to identify which questions are inclusion criteria and which are exclusion criteria. Only numbers should listed in the question number column.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 3c Inclusion/Exclusion Criteria Confirmation

| Unique<br>Patient<br>ID | Eligibility<br>confirmation | Eligibility<br>Confirmation<br>Date(DD-MM-<br>YYYY) | Eligibility<br>Re-confirmation | Eligibility<br>Re-confirmation<br>Date(DD-MM-YYYY) |
|---|---|---|---|---|
| xxxxx | xxxxx | DD-MM-YYYY | XXXXX | DD-MM-YYYY |
| XXXXX | XXXXX | DD-MM-YYYY | XXXXX | DD-MM-YYYY |
| XXXXX | XXXXX | DD-MM-YYYY | xxxxx | DD-MM-YYYY |

 ${\tt Code: S:\Services\setminus Immodulon\setminus IMM-101-008\setminus Analysis\setminus Development\setminus Code\setminus Listing 3c.sas \ ddmmmyy:hh:mm:ss.}$ 

 ${\tt Data: S:\Services\setminusImmodulon\setminusIMM-101-008\setminus xxxxx.sas7bdat}$ 

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Eligibility re-confirmation date is date of Day 0 (CRF page 11)

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

## Listing 4ai Melanoma Specific Medical History

| Unique<br>Patient<br>ID | Date of Initial Diagnosis of Current Presentation (DD-MM-YYYY) | Date of Excision of Primary Lesion (DD-MM-YYYY) | Date of Excision of Sentinel Node (DD-MM-YYYY) | Date of<br>Regional Lymph<br>Node Resection<br>(DD-MM-YYYY) | Date of Last<br>CT Scan<br>(DD-MM-YYYY) | Stage of<br>Disease | Primary<br>Lesion<br>Thickness<br>(T type) | Presence of<br>Lymph Node<br>Metastases<br>(N Type) |
|---|---|---|---|---|---|---|---|---|
| xxxxx | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | xxxxx | xxxxx | xxxxx |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | XXXXX |

Note: Dates have been listed where provided.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing4ai.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown/Not resected/Not excised/other specified text should be presented in the appropriate columns where applicable.

Note to programmer: Date of last CT scan is from CRF page 4: Disease and Treatment History

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

# Listing 4aii Melanoma Specific Medical History Continued

| | Ti | me (years) | since | | Lesion(s) details | | | | 3 |
|---|---|---|---|---|---|---|---|---|---|
| Unique | Initial | Excision | Excision | Regional | Presence | Melanoma | Longest | Shortest | Location |
| Patient | Diagnosis of | of | of | Lymph | of Current | Lesion | Diameter | Diameter | of Lesion |
| ID | Current | Primary | Sentinel | Node | Lesions | Number | (mm) | (mm) | |
| | Presentation | Lesion | Node | Resection | | | | | |
| XXXXX | XX | XX | XX | XX | XXXXX | 1 | X.XX | X.XX | XXXXX |
| | | | | | | 2 | X.XX | X.XX | XXXXX |
| | | | | | | 3 | X.XX | X.XX | XXXXX |
| | | | | | | 4 | X.XX | X.XX | XXXXX |
| XXXXX | XX | XX | XX | XX | XXXXX | 1 | X.XX | X.XX | XXXXX |
| | | | | | | 2 | X.XX | X.XX | XXXXX |

Note: Time (years) since variables are calculated from Day 0 + 1 and divided by 365.25.

Note: The screening assessment visible cutaneous lesions measurements were not recorded. Post screening assessment of lesions was not requested in the CRF.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing4aii.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Please add footnote if any 'time since' variables contain partial missing dates, see SAP section 8.2: Where day and month are not known for either date, calculation is based on year alone: Time since event (years) = (Year of Day 0 - Year of event) + 1/365.25.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Listing 4b
Significant Medical History since Completion of Study IMM-101-001

| Unique<br>Patient<br>ID | No<br>Significant<br>Medical<br>History | Body<br>system<br>Code* | Diagnosis | Preferred<br>Term | System<br>Organ<br>Class | Treatment | Start Date<br>(DD-MM-<br>YYYY) | Stop Date<br>(DD-MM-YYYY) | Anti-melanoma<br>Cancer Therapy |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | xxxxx | XXXXX | xxxxx | xxxxx | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |

Note: \*As recorded by the investigator

Note: Significant medical history includes all relevant anti-melanoma cancer therapy (radiotherapy, cancer surgery, chemotherapy, immunotherapy etc.) other than IMM-101 since finishing study IMM-101-001. Anti-melanoma cancer therapies are determined by the Sponsor's medical reviewer and flagged in the Anti-melanoma Cancer Therapy column.

Note: Preferred terms are coded using MedDRA version xx.x

Note: Ongoing is recorded as free text in the CRF where provided.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing4b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown should be presented in the appropriate date columns were applicable.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

Listing 5
Pre-Existing Injection Site Reaction(s) Assessed at Screening

| Unique<br>Patient<br>ID | Injection Site<br>Reaction Present | Counts Right<br>Deltoid | Counts Left<br>Deltoid | Do(es) The Local<br>Reaction(s) Affect<br>Daily Activities? | Comments<br>(where<br>applicable) |
|---|---|---|---|---|---|
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |
| XXXXX | XXXXX | XXXXX | XXXXX | xxxxx | XXXXX |

Note: Counts = Number of pre-existing injection site reactions present.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing5.sas ddmmmyy:hh:mm:ss

 ${\tt Data: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash xxxxx.sas7bdat}$ 

Note to programmer: Please update data footnote with appropriate file directory.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Listing 6
Screening Urine Pregnancy Test Results

| _ | Unique Patient ID | Result | Reason Test Not<br>Performed (if<br>applicable) |
|---|---|---|---|
| | xxxxx | XXXXX | xxxxx |
| | xxxxx | xxxxx | XXXXX |
| | xxxxx | XXXXX | XXXXX |
| | xxxxx | XXXXX | xxxxx |
| | xxxxx | xxxxx | XXXXX |
| | xxxxx | xxxxx | xxxxx |
| | xxxxx | xxxxx | ××××× |
| | AAAXX | AAAAX | AAXXX |
| | XXXXX | XXXXX | XXXXX |

Note: Test performed should be one of Yes, No, Not done or N/A (where N/A represents either males, or females who have had a hysterectomy)

 ${\tt Code: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash Analysis\backslash Development\backslash Code\backslash Listing 6.sas \ ddmmmyy:hh:mm:ss}$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Reason test not preformed is recorded in LBREASND.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y Analysis Population: Safety Population

> Listing 7 Disease and Treatment History at Screening

| Unique<br>Patient ID | Any medication within last 28 days ongoing or ceased? | Any IMM-101 administrations since patient completed Phase 1 study IMM-101- 001? | Significant or clinically relevant medical history since completing IMM-101-001? | History of severe local reaction following previous administrations of IMM-101? | Comments | Date of last CT scan<br>(DD-MM-YYYY) |
|---|---|---|---|---|---|---|
| XXXXX | XX | XX | xxxxx | XXXXX | XXXXX | DD-MM-YYYY |
| XXXXX | XX | XX | xxxxx | xxxxx | XXXXX | DD-MM-YYYY |
| XXXXX | XX | XX | xxxxx | xxxxx | XXXXX | DD-MM-YYYY |
| XXXXX | XX | XX | XXXXX | xxxxx | XXXXX | DD-MM-YYYY |
| xxxxx | XX | XX | XXXXX | xxxxx | xxxxx | DD-MM-YYYY |
| xxxxx | XX | XX | XXXXX | xxxxx | xxxxx | DD-MM-YYYY |
| xxxxx | XX | XX | XXXXX | xxxxx | xxxxx | DD-MM-YYYY |
| xxxxx | XX | XX | xxxxx | xxxxx | xxxxx | DD-MM-YYYY |

Note: Refer to Listing 4b for CRF page 7 comments.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing7.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: If unknown is recorded, for date of last CT scan, it should be included in the column were applicable.

Note to programmer: Date of last CT scan is from CRF page 8: Melanoma Specific History.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Listing 8a Previous Medications

| Unique<br>Patient ID | Previous<br>Medications<br>Taken is None | Reported<br>Name of Drug | Dose | Dose<br>Units | Indication | Start<br>Date<br>(DD-MM-<br>YYYY) | End Date<br>(DD-MM-<br>YYYY) | Was the<br>Mediation Taken<br>and Stopped<br>Before 14 days<br>Prior to Day 0? | Anti-melanoma<br>Cancer Therapy |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | x | xxxxx | | | xxxxx | DD-MM- | DD-MM- | X | |
| | | | X.XX | XX | | YYYY | YYYY | | |
| XXXXX | X | XXXXX | X.XX | | XXXXX | DD-MM- | DD-MM- | X | XXXXXXX |
| | | | | XX | | YYYY | YYYY | | |
| XXXXX | X | XXXXX | X.XX | | XXXXX | DD-MM- | DD-MM- | X | |
| | | | | XX | | YYYY | YYYY | | |

Note: Previous medications are all medications (prescription/non-prescription), including vitamins, drugs of abuse, and dietary supplements taken and stopped within 14 days prior to the end of screening procedures (i.e. Day 0). Any previous medications taken and stopped before 14 days prior to Day 0 have been flagged and included in the listing.

Note: Anti-melanoma cancer therapies are determined by the Sponsor's medical reviewer and flagged in the Anti-melanoma Cancer Therapy column.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing8a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown should be presented in the appropriate date columns were applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

## Listing 8b Concomitant Therapies

| Unique<br>Patient<br>ID | Reported Name<br>of Drug | Indication | Dose | Dose<br>Units | Dosing<br>Frequency | Start Date<br>(DD-MM-YYYY) | End Date<br>(DD-MM-YYYY) | Anti-melanoma<br>Cancer Therapy |
|---|---|---|---|---|---|---|---|---|
| XXXXX | xxxxx | XXXXX | x.xx | XX | xxxxx | DD-MM-YYYY | DD-MM-YYYY | XXXXXXX |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXXXXX |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |
| XXXXX | XXXXX | XXXXX | X.XX | XX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | |

Note: Concomitant Medications are all medications (prescription/non-prescription), including vitamins, and dietary supplements and surgical procedures ongoing or started on/after Day 0.

Note: Anti-melanoma cancer therapies are determined by the Sponsor's medical reviewer and flagged in the Anti-melanoma Cancer Therapy column.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing8b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Unknown should be presented in the appropriate date columns were applicable.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 9
Previous IMM-101 Administrations Since Completion of Study IMM-101-001

| Unique Patient<br>ID | Date of Last Administration of IMM-101 in Study IMM-101-001 (DD-MM-YYYY) | Administration Date of IMM-101 Since Completion of IMM-101-001 (DD-MM-YYYY) | Dose<br>(mg) | Injection<br>Site (R or<br>L Deltoid) |
|---|---|---|---|---|
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | X.XX | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | x.xx | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | X.XX | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | x.xx | XXXXX |
| XXXXX | DD-MM-YYYY | DD-MM-YYYY | X.XX | xxxxx |

Note: IMM-101 administrations since completion of IMM-101-001 were taken whilst patient was in Named Patient Programme and injection location was not recorded during this period.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing9.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: If date of administration is recorded as not known, present Unknown in place of date for the relevant dose.

Note to programmer: Date of last administration of IMM-101 in IMM-101-001 study should be displayed only once per patient.

S:\Services\Immodulon\IMM-101-008\SMF\SAP\IMM-101-008\_ SAPvFinal 1.1


## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

# Listing 10 On-Study IMM-101 Administration

| Unique<br>Patient<br>ID | Visit<br>Name/<br>Number | Visit Date | Date of Last<br>Dose of IMM-<br>101<br>(DD-MM-YYYY) | Have at Least 14 Days Passed Since Last Dose? | Time Elapsed Between This and Previous Dose (days) | Dose<br>Administered<br>(Y/N) | Dose<br>(mg) | Dose<br>Changed<br>From<br>Previous<br>Dose | Reason for<br>Dose<br>Reduction or<br>Delay (if<br>applicable) | Injection<br>Site |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | xx | x.xx | Х | xxxxx | xxxxx |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | x.xx | Х | xxxxx | xxxxx |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | Х | xxxxx | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | XXXXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | Х | XXXXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | XXXXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | xxxxx | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXX | XX | XX | X.XX | X | xxxxx | XXXXX |

Note: Time elapsed since previous dose (days) = (date of current dose - date of previous dose + 1).

Note: Dose changed from previous dose; I = increased, D = decreased (when compared with previous IMM-101 dose).

Note: Reasons for dose increases were also recorded in the CRF, as indicated.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing10.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Injection site should include right/left deltoid and upper/lower.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 11 On-Study Disease Assessment

| Unique<br>Patient ID | Visit<br>Name/Number | Visit Date<br>(DD-MM-YYYY) | Has a CT Scan been conducted since the last visit? (Y/N) | If yes, at the investigator's discretion, please indicate disease status compared to the last assessment | Comment (if applicable) |
|---|---|---|---|---|---|
| xxxxx | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | XX | XXXXX | xxxxx |
| XXXXX | XXXXX | DD-MM-YYYY | xx | xxxxx | xxxxx |

Note: Per protocol Investigator was asked to assess the presence of metastatic disease (if applicable) periodically following CT or MRI scan performed as routine standard of care.

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing11.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

## Listing 12 Adverse Events

| AE<br>No. | Reported<br>AE term | Preferred<br>Term | System<br>Organ<br>Class | Intensity<br>(CTCAE) | Seriousness<br>(N/Y) | Reason for<br>Seriousness/<br>Details if<br>other | Relationship<br>to Study<br>Drug | Start Date/Time<br>(DD-MM-YYYY<br>HH:MM) | End Date/Time (DD-MM-YYYY HH:MM) | Outco<br>me | Sequelae |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XX | xxxxx | xxxxx | xxxxx | xxxxx | XX | xxxxx | xxxxx | DD-MM-YYYY HH:MM | DD-MM-YYYY HH:MM | xxxxx | xxxxx |
| XX | XXXXX | XXXXX | xxxxx | XXXXX | XX | XXXXX | XXXXX | DD-MM-YYYY HH:MM | DD-MM-YYYY HH:MM | XXXXX | xxxxx |
| XX | XXXXX | XXXXX | XXXXX | XXXXX | XX | XXXXX | XXXXX | DD-MM-YYYY HH:MM | DD-MM-YYYY HH:MM | XXXXX | XXXXX |
| | No. xx xx xx xx xx xx xx | XX XXXXX XX XXXXX | No. AE term Term xx xxxxx xxxxx xx xxxxx xxxxx | No. AE term Term Organ Class xx xxxxx xxxxx xxxxx xx xxxxx xxxxx xxxxx | No. AE term Term Organ (CTCAE) xx xxxxx xxxxx xxxxx xx xxxxx xxxxx xxxxx | No. AE term Term Organ Class (CTCAE) (N/Y) xx xxxxx xxxxx xxxxx xxxxx xxxxx xx xx xxxxx xxxxx xxxxx xx xx xx xxxxx xxxxx xxxxx xx xx xxxxx xxxxx xx | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ Details if other xx xxxxx xxxxx xxxxx xxxxx xxxxx xx xxxxx xxxxx xxxxx xxxxx | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ other to Study Drug other xx xxxxx xxxxxx xxxxxx xxxxxx xxxxxx | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ other to Study (DD-MM-YYYY HH:MM) xx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM xx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ betails if other to Study (DD-MM-YYYY (DD-MM-YYYY HH:MM) (DD-MM-YYYY HH:MM) HH:MM) xx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx DD-MM-YYYY HH:MM DD-MM-YYYY HH:MM | No. AE term Term Organ (CTCAE) (N/Y) Seriousness/ to Study Drug HH:MM) HH:MM) xx xxxxx xxxxx xxxxx xxxxx xxxxx xxxxx xxxx |

Note: Treatment emergent AEs are all those reported during the study. Sequelae column also contains comments recorded in the sequelae field of the CRF.

Note: Preferred Term and System Organ Class are coded using MedDRA version x.xx.

Note: Common Toxicity Criteria for Adverse Events CTCAE code. 1. Mild, 2. Moderate, 3. Severe, 4. Life Threatening, 5. Death

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing12.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Where applicable, separate date from time using a space.

Note to Programmer: If Reason for seriousness is other please include reason/description.

Note to Programmer: Intensity should be occupied with text, the numeric CTCAE codes are provided in a note.

Note to programmer: Please add relevant version number in MedDRA note to reflect version used at time of coding.

Note to programmer: If necessary, break table over two pages with each new section of the table displaying Unique Patient ID, AE No., Reported AE term, Treatment Emergent, Preferred Term and System Organ Class.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

# Listing 13 On-Study Injection Site Reaction(s)

| Unique<br>Patient<br>ID | Visit<br>Name/<br>Number | Visit Date<br>(DD-MM-YYYY) | Date Last Dose of IMM-101 Administered (DD-MM-YYYY) | Is/are Injection Site Reaction(s) Visible From Previous Doses(s) of IMM-101? | Do(es) the Local Reaction(s) Affect Daily Activities? | Are Injection Site<br>Reactions Becoming<br>More Troublesome<br>With Repeated<br>Doses of IMM-101 | Wound Care<br>Required | Description<br>of Wound<br>Care<br>Provided |
|---|---|---|---|---|---|---|---|---|
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | XXXXX | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | xxxxx | XXXXX | XXXXX | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | xxxxx | XXXXX | xxxxx | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | xxxxx | XXX | XXXXX |
| XXXXX | XXXXX | DD-MM-YYYY | DD-MM-YYYY | XXXXX | XXXXX | XXXXX | XXX | xxxxx |

 ${\tt Code: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash Analysis\backslash Development\backslash Code\backslash Listing 13.sas \ ddmmmyy: hh:mm:ss} \\$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Listing 14
Concomitant Medication and Adverse Event Checks

| Unique<br>Patient ID | Visit<br>Name/Number | Visit<br>Date<br>(DD-MM-YYYY) | Any medication (prescription or non-prescription) started or ceased since the last dose of IMM-101? (Y/N/Unknown) | Other than a local reaction, did the patient have any concurrent sign(s), symptoms(s), and or disease(s)? (Y/N) |
|---|---|---|---|---|
| xxxxx | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | XX | DD-MM-YYYY | xxxxx | xxxxx |

Note: UK, U = Unknown.

 ${\tt Code: S:\Services\setminus Immodulon\setminus IMM-101-008\setminus Analysis\setminus Development\setminus Code\setminus Listing 14.sas \ ddmmmyy: hh:mm:ss} \\$ 

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y

Analysis Population: Safety Population

Listing 15 Study Visits and Visit Checklists

| Unique Patient<br>ID | Visit<br>Name/Number | Visit Date (DD-MM-YYYY) | Number of weeks<br>elapsed since last<br>visit (where<br>applicable) | Checklist Item | Completed (Y/N) |
|---|---|---|---|---|---|
| xxxxx | xxxxx | DD-MM-YYYY | XX | xxxxx | XX |
| xxxxx | xxxxx | DD-MM-YYYY | XX | xxxxx | XX |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing15.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Include Date of Consent for patient transfer to Site 2, date of first visit at Site 2 and nominal visit number according to CRF entries, in chronological order in the listing (see Immodulon file note FN47).

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

Note to programmer: All visits should be listed. Checklist items text to be stated in full. If text too long, add a key on separate listing 15a or similar.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 16
Blood Sample for Immunological Markers

| Unique Patient ID | Visit Name/<br>Number | Visit Date<br>(DD-MM-YYYY) | Blood Sample Taken?<br>(Y/N) | Volume (mL) |
|---|---|---|---|---|
| xxxxx | XXXXX | DD-MM-YYYY | XX | XX.X |
| XXXXX | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |
| XXXXX | XXXXX | DD-MM-YYYY | xx | XX.X |
| xxxxx | XXXXX | DD-MM-YYYY | xx | XX.X |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing16.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Visit Name/Number should be one of Screening, Day 0 or Routine Visit xx.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008 Page x of y

Analysis Population: Safety Population

# Listing 17 Post-Study Long Term Survival Status

| Unique Patient<br>ID | Date of Consent For<br>Data Collection | Date of Assessment<br>of Status<br>(DD-MM-YYYY) | Survival Status | If Death, Date of Death (DD-MM-YYYY) | If Death,<br>Cause of<br>Death | Investigator<br>Signature<br>Date<br>(DD-MM-YYYY) |
|---|---|---|---|---|---|---|
| xxxxx | XXXXX | DD-MM-YYYY | xxxx | DD-MM-YYYY | xxxxx | xxxxx |
| XXXXX | xxxxx | DD-MM-YYYY | xxxx | DD-MM-YYYY | XXXXX | XXXXX |

 $\label{lem:code:s:Services} Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing17.sas \ ddmmmyy:hh:mm:ss$ 

 ${\tt Data: S:\Services\backslash Immodulon\backslash IMM-101-008\backslash xxxxx.sas7bdat}$ 

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Data is recorded on Post-study Survival Status CRF, with multiple rows per patient (depending on number of occasions long term survival status is assessed).

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Listing 18
Additional Comments Recorded

| Unique Patient<br>ID | Related Domain | Visit at which comment recorded | Date of Visit<br>(DD-MM-YYYY) | Associated Variable | Comment |
|---|---|---|---|---|---|
| xxxxx | XXXX | xxxxx | DD-MM-YYYY | xxxx | XXXXX |
| XXXXX | xxxx | XXXXX | DD-MM-YYYY | XXXX | XXXXX |

Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Listing18.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: Data is recorded as free text comments on the CRF.

Note to programmer: Please sort the listing by patient ID and related domain.

Note to programmer: For any comment relating to AEs, please put the 'AE xx:' in front of the comment.

# **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y Analysis Population: Safety Population

Figure 1a Panel Plot of On-Study IMM-101 Doses by Patient



Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Figure1a.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: A plot for each patient should be produced (with patient number in the subtitle for each plot) and all plots should be displayed in a panel plot (2x5). Each dose should be marked on the line plot by an 'X' or similar.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Page x of y Analysis Population: Safety Population

Figure 1b All IMM-101 Dosing Administrations (IMM-101-001 and IMM-101-008 Combined)



Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\ Figure1b.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\ xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to programmer: A plot for each patient should be produced (with patient number in the subtitle for each plot) and all plots should be displayed in a panel plot (2x5 landscape format). Each dose should be marked on the line plot by an 'X' or similar. Standard axes should be used across the plots.

## **Exploristics Limited**

Identifier: EXP12002

Clinical Study Identifier: IMM-101-008

Final Analysis

Protocol: IMM-101-008

Analysis Population: Safety Population

Page x of y

Figure 2
Kaplan Meier Curve of Overall Survival



Code: S:\Services\Immodulon\IMM-101-008\Analysis\Development\Code\Figure2.sas ddmmmyy:hh:mm:ss

Data: S:\Services\Immodulon\IMM-101-008\xxxxx.sas7bdat

Note to programmer: Please update data footnote with appropriate file directory.

Note to Programmer: Add Label along X-axis: Time (Years) after Day 0 date (X-axis range according to the time to event). Add Y-axis Proportion Alive. Include markers for withdrawn/censored patients.